# Statistical Analysis Plan

Cetero Research Protocol No. CTJK09001 Theracos, Inc. Protocol No. THR-1442-C-402

A Phase II, four-week, multi-center, double-blind, placebo-controlled parallel group study to evaluate the safety and efficacy of EGT0001442 in subjects with type 2 Diabetes Mellitus with an ascending dose safety and pharmacokinetic evaluation period

Cetero Research 4520 Dixie Road Mississauga, Ontario, L4W 1N2 Canada

> 17-May-2010 Final Version 1.0

| Written By: | | |
|--------------|--------------------------------|------|
| | Jianhua Liu, M.Sc. | Date |
| | Manager Biostatistics | |
| | Cetero Research | |
| Approved by: | | |
| ,, | Pina D'Angelo, M.Sc. | Date |
| | Director Biostatistics & PK/PD | |
| | Cetero Research | |
| | Yuan-Di Halvorsen, Ph.D. | Date |
| | Clinical Project Leader | |
| | Theracos, Inc. | |

# Statistical Analysis Plan

Cetero Research Protocol No. CTJK09001 Theracos, Inc. Protocol No. THR-1442-C-402

A Phase II, four-week, multi-center, double-blind, placebo-controlled parallel group study to evaluate the safety and efficacy of EGT0001442 in subjects with type 2 Diabetes Mellitus with an ascending dose safety and pharmacokinetic evaluation period

Cetero Research 4520 Dixie Road Mississauga, Ontario, L4W 1N2 Canada

> 17-May-2010 Final Version 1.0

| Written By: | 7 Siv | 25-May-2010 |
|---|---|---|
| • | Jianhua Liu, M.Sc.<br>Manager Biostatistics<br>Cetero Research | Date |
| Approved by: | Pina D'Angelo, M.Sc. Director Biostatistics & PK/PD Cetero Research | 25 - MAY - 2016<br>Date |
| | Yuan-Di Halvorsen, Ph.D. Clinical Project Leader Theracos, Inc. | May 25, 2010 Date |

# LIST OF ABBREVIATIONS AND DEFINITIONS OF TERMS

AE adverse event

ANOVA analysis of variance

ATC the anatomic therapeutic chemical classification

AUC area under the curve

AUC<sub>0-t</sub> area under the plasma concentration-time curve from time 0 to time t

(time of last quantifiable plasma concentration)

AUC<sub>0-inf</sub> area under the plasma concentration-time curve from time 0 to infinity

AUC<sub>0-24</sub> area under the plasma concentration-time curve from time 0 to 24 h

BMI body mass index

CI confidence interval

CL/F the apparent total body clearance

C<sub>max</sub> maximum observed plasma concentration

CRF case report form

CV coefficient of variation

DSMB data and safety monitoring board

ECG electrocardiogram

FDA food and drug administration

FPG fasting plasma glucose

GCP good clinical practice

HbA1c glycated hemoglobin

ICH international conference on harmonisation

ITT intent-to-treat

Kel terminal phase rate constant

MedDRA medical dictionary for regulatory activities

PK pharmacokinetics

PP per protocol

SAE serious adverse event

SAP statistical analysis plan

SD standard deviation

SMBG self monitored blood glucose

TEAE treatment emergent adverse event

Thalf apparent terminal half life

 $T_{\text{max}}$  time of observed maximum plasma concentration

UGE0-24 urinary glucose excretion from 0 to 24 h post dose

 $V_z/F$  the apparent total volume of distribution

# **Table of Contents**

| List of Abbreviations and Definitions of Terms | 2 |
|---|---|
| 1. INTRODUCTION | 8 |
| 2. OBJECTIVES | 8 |
| 3. OVERALL STUDY DESIGN AND PLAN | 9 |
| 4. TREATMENT ADMINISTERED | |
| 5. BLINDING | |
| 6. METHOD OF ASSIGNING SUBJECTS TO TREATMENT GROUPS | 11 |
| 7. SAMPLE SIZE | |
| 8. ANALYSIS POPULATIONS | |
| 9. STUDY ENDPOINTS | |
| 10. STATISTICAL METHODS | |
| 10.1 Baseline Characteristics | |
| 10.1.1 Demographics and Baseline Characteristics | |
| 10.1.2 Medical History | |
| 10.1.3 Inclusion/Exclusion Criteria and Exceptions | |
| 10.1.4 Urine Drug Screen | |
| 10.2 Primary Analysis | |
| 10.3 Secondary Analyses | |
| 10.4 Safety Analysis | |
| 10.4.1 Adverse Event Analysis | |
| 10.4.2 Clinical Laboratory Tests | |
| 10.4.3 Concomitant Medication | |
| 10.4.4 FPG, Vital Signs, SMBG record, and ECG Parameters | |
| 10.4.5 Physical Exam | |
| 10.5 PK Assessments | |
| 10.6 Exploratory Analysis of the Post-prandial Blood Glucose | 19 |
| 10.7 Interim Analysis | |
| 10.8 Missing Data | |
| 10.9 Multiple Comparisons | |
| 11. TABLE, LISTING AND FIGURE SHELLS | 20 |
| , | |
| Tables: | |
| Table 14.1.1 Disposition of Subjects (Double-blind Segment) | 22 |
| Table 14.1.2 Disposition of Subjects (Dose Escalation Segment) | 23 |
| Table 14.1.3 Summary of Demographics (Double-blind Segment) | 24 |
| Table 14.1.4 Summary of Demographics (Dose Escalation Segment) | |
| Table 14.2.1 Primary Efficacy Analysis: Descriptive Summary of Fasting Plasma Glucose | |
| from Baseline to End of Treatment Double-blind Segment Intent-to-Treat Analysis Set | 28 |
| Table 14.2.2 Primary Efficacy Analysis: ANCOVA Results on Mean Change in FPG from | |
| Baseline to End of Treatment Double-blind Segment Intent-to-Treat Analysis Set | 29 |
| Table 14.2.3 Descriptive Summary of Fasting Plasma Glucose from Baseline to End of | |
| Treatment Double-blind Segment Per-Protocol Analysis Set | 30 |
| Table 14.2.4 ANCOVA Results on Mean Change in FPG from Baseline to End of | |
| Treatment Double-blind Segment Per-Protocol Analysis Set | 30 |
| Table 14.2.5 Descriptive Summary of Fasting Plasma Glucose from End of Treatment to | |
| Post Treatment Double-blind Segment Intent-to-Treat Analysis Set | 31 |

| Table 14.2.6 ANCOVA Results on Mean Change in FPG from End of Treatment to Post | |
|---|---|
| Treatment Double-blind Segment Intent-to-Treat Analysis Set | . 32 |
| Table 14.2.7 Descriptive Summary of Change in Body Weight from Baseline to Day 29 | |
| Double-blind Segment Intent-to-Treat Analysis Set | . 33 |
| Table 14.2.8 ANCOVA Results on Mean Change in Body Weight from Baseline to Day 29 | |
| Double-blind Segment Intent-to-Treat Analysis Set | . 34 |
| Table 14.2.9 Descriptive Summary of Change in HbA1c from Baseline to Day 29 Double- | |
| blind Segment Intent-to-Treat Analysis Set | . 35 |
| Table 14.2.10 ANCOVA Results on Mean Change in HbA1c from Baseline to Day 29 | |
| Double-blind Segment Intent-to-Treat Analysis Set | . 36 |
| Table 14.2.11 Descriptive Summary of Change in 24 h UGE from Baseline to Day 28 | |
| Double-blind Segment Intent-to-Treat Analysis Set | . 37 |
| Table 14.2.12 ANCOVA Results on Mean Change in 24 h UGE from Baseline to Day 28 | . 57 |
| · | 20 |
| Double-blind Segment Intent-to-Treat Analysis Set | . 38 |
| Table 14.2.13 Summary of Plasma Concentrations of EGT0001442 (ng/mL) Dose | 20 |
| Escalation Segment | . 39 |
| Table 14.2.14 Summary of Pharmacokinetic Parameters of EGT0001442 Dose Escalation | |
| Segment | . 40 |
| Table 14.2.15 Summary of Post Prandial Blood Glucose (mg/dL) in Change from Day 0 to | |
| Day 2 Dose Escalation Segment | . 41 |
| Table 14.2.16 Summary of Post Prandial Blood Glucose in AUC Dose Escalation | |
| Segment | . 42 |
| Table 14.3.1.1 Summary of TEAEs Double-blind Segment Double-blind Safety Analysis | |
| Set | . 43 |
| Table 14.3.1.2 Summary of TEAEs Dose Escalation Segment Dose Escalation Safety | |
| Analysis Set | . 44 |
| Table 14.3.1.3 Summary of TEAEs by System Organ Class, Preferred Term and | |
| Treatment Group Double-blind Segment Double-blind Safety Analysis Set | . 45 |
| Table 14.3.1.4 Summary of Drug-related TEAEs by System Organ Class, Preferred Term | |
| and Treatment Group Double-blind Segment Double-blind Safety Analysis Set | . 46 |
| Table 14.3.1.5 Summary of TEAEs Leading to Study Discontinuation by System Organ | |
| Class, Preferred Term and Treatment Group Double-blind Segment Double-blind | |
| Safety Analysis Set | . 46 |
| Table 14.3.1.6 Summary of Serious TEAEs by System Organ Class, Preferred Term and | |
| Treatment Group Double-blind Segment Double-blind Safety Analysis Set | . 46 |
| Table 14.3.1.7 Summary of TEAEs by System Organ Class, Preferred Term and Dose | |
| | 47 |
| Table 14.3.1.8 Summary of Drug-related TEAEs by System Organ Class, Preferred Term | |
| and Dose Group Dose Escalation Segment Dose Escalation Safety Analysis Set | 48 |
| Table 14.3.1.9 Summary of TEAEs Leading to Study Discontinuation by System Organ | |
| Class, Preferred Term and Dose Group Dose Escalation Segment Dose Escalation | |
| | . 48 |
| Safety Analysis SetTable 14.3.1.10 Summary of Serious TEAEs by System Organ Class, Preferred Term and | +0 |
| | . 48 |
| · | 40 |
| Table 14.3.1.11 Summary of TEAEs by Maximum Severity Double-blind Segment | 10 |
| Double-blind Safety Analysis Set | . 49 |
| Table 14.3.1.12 Summary of TEAEs by Maximum Severity Dose Escalation Segment | |
| | . 50 |
| Table 14.3.1.13 Clinical Laboratory Evaluations in Biochemistry (Observed Values) | _ |
| Double-blind Seament Double-blind Safety Analysis Set | . 51 |

| Table 14.3.1.14 Clinical Laboratory Evaluations in Change from Baseline in Biochemistry | |
|---|---|
| Double-blind Segment Double-blind Safety Analysis Set | 52 |
| Table 14.3.1.15 Biochemistry Laboratory Shift Table Double-blind Segment Double-blind Safety Analysis Set | ı<br>53 |
| Table 14.3.1.16 Clinical Laboratory Evaluations in Hematology (Observed Values) | 55 |
| Double-blind Segment Double-blind Safety Analysis Set | 54 |
| Table 14.3.1.17 Clinical Laboratory Evaluations in Change from Baseline in Hematology | 57 |
| Double-blind Segment Double-blind Safety Analysis Set | 54 |
| Table 14.3.1.18 Hematology Laboratory Shift Table Double-blind Segment Double-blind | 0- |
| Safety Analysis Set | 54 |
| Table 14.3.1.19 Clinical Laboratory Evaluations in Urinalysis (Observed Values) Double- | |
| blind Segment Double-blind Safety Analysis Set | 54 |
| Table 14.3.1.20 Clinical Laboratory Evaluations in Change from Baseline in Urinalysis | |
| Double-blind Segment Double-blind Safety Analysis Set | 54 |
| Table 14.3.1.21 Urinalysis Laboratory Shift Table Double-blind Segment Double-blind | |
| Safety Analysis Set | 55 |
| Table 14.3.1.22 Clinical Laboratory Evaluations in Biochemistry (Observed Values) Dose | |
| Escalation Segment Dose Escalation Safety Analysis Set | 56 |
| Table 14.3.1.23 Clinical Laboratory Evaluations in Hematology (Observed Values) Dose | |
| Escalation Segment Dose Escalation Safety Analysis Set | 57 |
| Table 14.3.1.24 Clinical Laboratory Evaluations in Urinalysis (Observed Values) Dose | |
| Escalation Segment Dose Escalation Safety Analysis Set | 57 |
| Table 14.3.1.25 Summary of Vital Signs (Observed Values) Double-blind Segment | |
| Double-blind Safety Analysis Set | 58 |
| Table 14.3.1.26 Summary of Vital Signs in Change from Baseline Double-blind Segment | |
| Double-blind Safety Analysis Set | 59 |
| Table 14.3.1.27 Summary of Vital Signs (Observed Values) Dose Escalation Segment | |
| Dose Escalation Safety Analysis Set | 60 |
| Table 14.3.1.28 Summary of 12-Lead ECG (Observed Values) Double-blind Segment | |
| Double-blind Safety Analysis Set | 61 |
| Table 14.3.1.29 Summary of 12-Lead ECG in Change from Baseline Double-blind | 60 |
| | 62 |
| Table 14.3.1.30 Summary of 12-Lead ECG (Observed Values) Dose Escalation Segment Dose Escalation Safety Analysis Set | 63 |
| Table 14.3.1.31 Summary of Fasting Plasma Glucose by Visit (Observed Values) Double | |
| blind Segment Double-blind Safety Analysis Set | |
| Table 14.3.1.32 Summary of Concomitant Medication Double-blind Segment Double- | 0- |
| blind Safety Analysis Set | 65 |
| Table 14.3.1.33 Summary of Concomitant Medication Dose Escalation Segment Dose | |
| Escalation Safety Analysis Set | . 66 |
| <u>Listings:</u> | |
| <del></del> | |
| Listing 16.2.1 Subject Disposition | 68 |
| Listing 16.2.2 Protocol Deviations | |
| Listing 16.2.3 Subjects Excluded from the Efficacy Analysis (Double-blind Segment) | |
| Listing 16.2.4.1 Demographics | 71 |
| Listing 16.2.4.2 Medical History | |
| Listing 16.2.4.3 Prior and Concomitant Medication | |
| Listing 16.2.4.4 Inclusion/Exclusion Criteria and Exceptions | |
| Listing 16.2.4.5 Urine Drug Screen | 75 |

| Listing 16.2.5 Study Drug Administration | . 76 |
|---|---|
| Listing 16.2.6.1 Fasting Plasma Glucose (mg/dL) | . 77 |
| Listing 16.2.6.2 Weight | . 78 |
| Listing 16.2.6.3 Glycated Hemoglobin A1 (HbA1c) (%) | . 79 |
| Listing 16.2.6.4 24 h UGE (g/day) | |
| Listing 16.2.6.5 Blood (PK) Sample Collection (Dose Escalation Segment) | . 81 |
| Listing 16.2.6.6 Post Prandial Blood Glucose (mg/dL) (Dose Escalation Segment) | |
| Listing 16.2.7.1 Treatment Emergent Adverse Events | . 83 |
| Listing 16.2.7.2 Drug-related Treatment Emergent Adverse Events | . 84 |
| Listing 16.2.7.3 Serious Treatment Emergent Adverse Events | . 84 |
| Listing 16.2.7.4 Treatment Emergent Adverse Events Leading to Study Discontinuation | . 84 |
| Listing 16.2.7.5 Cardiovascular Treatment Emergent Adverse Events | |
| Listing 16.2.7.6 Pre-treatment Adverse Events | |
| Listing 16.2.7.7 Adverse Events during Washout Period | . 86 |
| Listing 16.2.8.1 Clinical Laboratory Test Results in Biochemistry | |
| Listing 16.2.8.2 Clinical Laboratory Test Results in Hematology | . 88 |
| Listing 16.2.8.3 Clinical Laboratory Test Results in Urinalysis | |
| Listing 16.2.8.4 Vital Signs | . 89 |
| Listing 16.2.8.5 12-Lead ECG | . 90 |
| Listing 16.2.8.6 Self Monitored Blood Glucose (SMBG) | . 91 |
| Listing 16.2.8.7 Physical Examination | . 92 |
| <u>Figures:</u> | |
| Figure 14.2.1 Fasting Plasma Glucose (mean± SE) - Double-blind Segment | 04 |
| Figure 14.2.2 Fasting Plasma Glucose in Change from Baseline (mean± SE) - Double- | . 9 <del>4</del> |
| blind Segment | 05 |
| Figure 14.2.3 Body Weight (mean± SE) - Double-blind Segment | |
| Figure 14.2.4 Body Weight in Change from Baseline (mean± SE) - Double-blind Segment. | |
| Figure 14.2.5 HbA1c (mean± SE) - Double-blind Segment | . 90 |
| Figure 14.2.6 24h UGE (mean± SE) - Double-blind Segment | |
| Figure 14.2.7 Mean Plasma Concentration for EGT0001442 (ng/mL) - Dose Escalation | . 30 |
| SegmentSegment | an |
| Figure 14.2.8 Individual Plasma Concentration for EGT0001442 (ng/mL) - Dose Escalation | . ฮฮ<br>า |
| · | 100 |

# **Statistical Analysis Plan**

#### 1. INTRODUCTION

This SAP is based on the final Protocol THR-1442-C-402 Amendment 2 dated 23 February 2010. The SAP provides details on the planned statistical methodology for analysis of the study data. The SAP also outlines the statistical programming specifications for the tables, listings and figures.

This SAP describes the study endpoints, derived variables, anticipated data transformations and manipulations, and other details of the analyses not provided in the study protocol. This SAP therefore outlines in detail all other aspects pertaining to the planned analyses and presentations for this study.

The following documents were reviewed in preparation of this SAP:

- Clinical Research Protocol final Protocol THR-1442-C-402 Amendment 1 dated 23 February 2010
- Case report forms (CRFs) issued on 22 March 2010: R09-0980 (THR-1442-C-402) eCRF Template - Insubject V1.2.pdf and R09-0980 (THR-1442-C-402) eCRF Template - Outsubject V1.2.pdf
- ICH Guidance on Statistical Principles for Clinical Trials.

The reader of this SAP is encouraged to also read the clinical protocol for details on the conduct of this study, and the operational aspects of clinical assessments and timing for completing a subject in this study.

#### 2. OBJECTIVES

#### Primary Objectives:

The primary objectives of this study are:

- To determine the effect of EGT0001442 on fasting plasma glucose (FPG) at the end of 4 weeks of treatment.
- To assess the pharmacokinetics and safety and tolerability of EGT0001442 at four dose levels in diabetic subjects given the drug daily for 4 weeks.

# **Secondary Objectives:**

- To determine changes in body weight at week 4 from baseline.
- To determine changes in HbA1c at week 4 compared to baseline.
- To determine changes in FPG following cessation of treatment
- To determine the pharmacodynamics of EGT0001442 by urinary glucose excretion (UGE) in diabetic subjects on day 0, day 1 and day 28.

#### PK Objective:

To determine the pharmacokinetics of EGT0001442 in diabetic subjects

#### Exploratory Objective:

 To measure changes in post-prandial blood glucose from baseline to day 2 in the 20 subjects in the dose escalation segment of the trial while they remain supervised in the clinic.

#### 3. OVERALL STUDY DESIGN AND PLAN

EGT0001442 is an experimental agent being developed by Theracos Inc. for the treatment of type 2 diabetes. EGT0001442 is a selective inhibitor of human sodium glucose cotransporter 2 (SGLT2). A first-in-human study and a subsequent phase I study in diabetic subjects have previously evaluated the safety and tolerability of EGT0001442 (as proline cocrystal) up to a dose of 100 mg/d for 14 days (150 mg/d of cocrystal) in healthy volunteers or as a single dose of 100 mg (150 mg of cocrystal) in diabetic subjects. This trial is the first to expose human subjects to EGT0001442 as a single agent (i.e., not as proline cocrystal) and is conducted at dose levels of 5, 10, 20 and 50 mg per day, or placebo, in two segments.

The first segment is a single center, open labeled pharmacokinetic 3 day insubject study with a 25 day outsubject continuation, intended to assess any significant changes in the exposure to EGT0001442 when delivered by single agent crystal compared to proline cocrystal. The similar solubility and dissolution rate of the two formulations of EGT0001442 suggest that significant differences in exposure compared to those observed following proline cocrystal administration are unlikely. However a drug and safety monitoring board will review the outcomes and pharmacokinetic data to determine if the pharmacokinetic profile will result in the mean  $C_{\text{max}}$  or  $AUC_{0-24}$  exceeding the NOAEL in male rats (the limiting sex and species derived from 28 day repeat dosing studies).

The second segment of the proposed clinical evaluation is a multicenter, placebo-controlled, five-arm parallel group, double-blind, randomized clinical trial of 28 day duration conducted in an outsubject population. EGT0001442 delivered at dose levels of 5, 10, 20 and 50 mg per day, or placebo, is administered to approximately 25 subjects per dose for a period of 28 days followed by a 14 day follow-up period.

The primary objective of the second segment is to evaluate the efficacy of EGT0001442 in the treatment of type 2 diabetes mellitus. Approximately 125 subjects will be randomly assigned to receive EGT0001442 at 5, 10, 20, or 50 mg/day or placebo with an equal number of subjects per group.

The primary efficacy end point is the assessment of the effect of EGT0001442 on fasting plasma glucose (FPG) after 4 weeks on treatment compared to baseline FPG values. The secondary efficacy end points include:

- Changes in body weight at week 4 from baseline
- Changes in HbA1c at week 4 compared to baseline
- Change in FPG following cessation of treatment
- Pharmacodynamic effects of EGT0001442 on urinary glucose excretion (UGE) in

diabetic subjects on day 0 (baseline), day 1 and day 28.

Safety of EGT0001442 will be evaluated by assessment of adverse events and concomitant medication records, hematology and blood chemistry laboratory results, cardiovascular events, electrocardiograms (ECG), urine electrolytes and urinalysis.

PK parameters will be evaluated in the 20 subjects in the dose escalation segment. An exploratory analysis of changes in post-prandial blood glucose on day 0 and day 2 while in-clinic from subjects in the dose escalation segment will also be conducted.

#### 4. TREATMENT ADMINISTERED

In the open labeled, dose escalation segment, subjects will take one of the 5 mg, one of the 10 mg, two of the 10 mg, or two of the 25 mg EGT0001442 capsules daily in the 5, 10, 20, or 50 mg cohort.

In the outsubject randomization segment, the following treatments will be administered:

| Treatment group | Placebo<br>capsule /day | | 0001442<br>ules /day<br>10 | 25 | Total #<br>capsules/day |
|---|---|---|---|---|---|
| 5 mg EGT0001442 | 1 | 1 | | | 2 |
| 10 mg EGT0001442 | 1 | | 1 | | 2 |
| 20 mg EGT0001442 | | | 2 | | 2 |
| 50 mg EGT0001442 | | | | 2 | 2 |
| Placebo | 2 | | | | 2 |

Table 1. EGT0001442 or placebo treatments

During the dose escalation segment of the study, the study drug will be administered orally to subjects in the upright position with approximately 200 mL of water between 07:00 h and 10:00 h, following a minimum of a 10 h overnight fast. During fasting, no fluids will be taken in the two hours prior to drug administration. The capsules will be swallowed without chewing. Breakfast will be given 0.5 h after dosing. Administration of all study medications will be supervised. After drug administration, a hand and mouth inspection will take place.

In the outsubject setting, subjects will be instructed to self administer one capsule from each of the two bottles prior to breakfast once daily for 25 or 28 days, respectively, and complete the dosing log. Taking the study medication with a glass of water is recommended.

#### 5. BLINDING

The dose escalation segment of the study will be open labeled. In the randomization segment, the study drug will be blinded to the sponsor, investigators, the study coordinator, study subjects, and pharmacist. Upon randomization, each subject will receive a subject randomization number and a drug kit number assigned to the subject.

The dosing information will remain blinded to all of the study team until the last subject has completed the last follow up visit and the database has been locked. A designated statistician that will provide safety data upon request from the DSMB will be allowed to receive unblinded data.

To manage the safety monitoring and maintain blinding of the treatment, there will be an unblinded study staff who will review the FPG data and alert the investigator and essential study staff if glucose is below 2.8 mmol/L (50 mg/dL), 3.9 mmol/L (70 mg/dL), or above 12 mmol/L (216 mg/dL), 15 mmol/L (270 mg/dL) or 16.7 mmol/L (300 mg/dL). The actual numerical values of the FPG will remain blinded to all study personnel and subjects unless clinically indicated, as outlined in section 5.4.

The investigator will also receive a sealed envelope for each subject containing a description of the dispensed medication. The envelope can be opened only if knowledge of the test substance is needed to manage the subject's condition. If opened, the date of opening and the reason for opening must be written on the envelope. At the conclusion of the study, all envelopes must be returned to the Sponsor. These will be checked to ensure that the seals had not been broken, unless warranted by the occurrence of the events mentioned above. If unblinding occurs, the time and reason for unblinding will be recorded on the CRF and the sponsor must be notified within 24 h.

#### 6. METHOD OF ASSIGNING SUBJECTS TO TREATMENT GROUPS

The dose escalation segment of the study will be open labeled. Study drug will be provided to the site pharmacist in bottles of 30 capsules. The pharmacist will dispense the study drug to the subjects.

In the randomization segment, eligible subjects who complete the 15 ± 2 day washout period to verify eligibility for the study and stability of their diabetes will be randomized to receive EGT0001442 or placebo according to a randomization code generated by the Pharmacometric Department of the contract research organization (CRO). Approximately 125 subjects will be randomly assigned to a treatment group within each treatment center to control for any potential bias due to center. Subjects are assigned to placebo or EGT0001442 at doses of 5, 10, 20, or 50 mg/day in a 1:1:1:1:1 ratio. Randomization will be stratified by study center. Completion of a block of 5 will initiate the assignment of a new random block and the process will continue until all subjects are enrolled. This randomization protocol is designed to balance experimental treatments within each center.

The Outsubject Segment of this study will be conducted at multiple investigative sites and will likely involve variable numbers of subjects at each site. Enrollment will be on a competitive basis but will be capped at 40% of the total randomized subjects (50 subjects) from one center.

## 7. SAMPLE SIZE

The efficacy pairwise null and alternative hypotheses to be assessed are as follows:

$$H_{0i}$$
:  $\mu_i = \mu_P$   
VS.  
 $H_{1i}$ :  $\mu_i \neq \mu_P$ 

where  $\mu_i$  = the mean change in FPG from baseline to week 4 for dose i (i = 5, 10, 20 or 50 mg/day of EGT0001442) and  $\mu_P$  = the mean change in FPG from baseline to week 4 for placebo. The test of each pairwise null hypothesis will be carried out at the two-sided 0.05 level of significance; no adjustment for multiple comparisons will be made.

The sample size of 25 subjects per group was calculated based on the following assumptions:

- 1. Baseline mean (± standard deviation) FPG is 190 (± 40) mg/dL for each dose group;
- 2. The active doses will decrease FPG on average by 25 (± 25) mg/dL from baseline to day 28
- 3. The placebo will not experience a substantive average decrease in mean FPG from baseline to day 28; the standard deviation of the change in mean FPG from baseline to day 28 is assumed conservatively to be 25 (same standard deviation as for active doses).
- 4. The two-sided significance level for each pairwise hypothesis is 0.05.

Under the above assumptions, an evaluable sample size of 22 evaluable subjects per treatment arm yields approximately 90% power that at least one dose will be found to be significantly different from placebo. A sample size of 25 subjects per treatment arm will be enrolled to account for any subject lost-to-follow-up.

#### 8. ANALYSIS POPULATIONS

#### Intent-to-Treat Analysis Set:

All randomized subjects in segment 2 of the study. This is the analysis set on which efficacy endpoints will be evaluated. All subjects will be analyzed according to the treatment to which they were randomized. The Intent-to-Treat Analysis Set will be used to perform the efficacy analysis for the double-blind segment only.

#### Per-Protocol Analysis Set:

The subset of subjects from the Intent-to-Treat analysis set that received at least 24 doses of study drug to which they were randomized, did not miss more than one dose in the last week of study medication, did not have any major protocol deviations and were measured for FPG visit with confirmed ≥10 hour fast at the day 27 and day 29 visits within the specified visit window. Subjects who stopped treatment due to rescue medication are also included in the analysis set. All subjects will be analyzed according to the treatment received.

The Per-Protocol Analysis Set will be evaluated only for primary efficacy to confirm results from the Intent-to-Treat Analysis Set. The final subject evaluability will be performed prior to breaking treatment codes and locking the database.

#### Double-blind Safety Analysis Set:

All randomized subjects who receive at least one dose of treatment during the randomization segment. Subjects will be analyzed according to the treatment received. The Double-blind Safety Analysis Set will be used to perform safety assessments for the double-blind segment.

#### Dose-Escalation Safety Analysis Set:

All subjects who receive at least one dose of treatment during the dose escalation segment of the study. Subjects will be analyzed according to the treatment received.

The Dose-Escalation Safety Analysis Set will be used to perform safety assessments for the open-label dose escalation segment.

#### 9. STUDY ENDPOINTS

#### Primary Efficacy Endpoint

The primary efficacy endpoint is change in FPG.

# Secondary Efficacy Endpoints

- Change in body weight from baseline to day 29
- Change in HbA1c from baseline to day 29.
- Change in FPG from cessation of treatment (days 27/29 to days 41/43).
- 24 h UGE on day 0, day 1 and day 28

#### **Primary Safety Endpoints**

- Adverse events
- Clinical and laboratory variables
- Concomitant medication
- FPG, Vital signs, SMBG record, and ECG parameters

#### 10. STATISTICAL METHODS

Data will be summarized with respect to demographic and baseline characteristics, efficacy variables and safety variables.

Summary statistics will include the mean, N, standard deviation, median, minimum, and maximum values for continuous variables, and frequencies and percentages for categorical variables.

If not otherwise specified, all statistical analyses will be two-sided and the Type I (alpha) error is fixed at the 5% level.

#### 10.1 Baseline Characteristics

# 10.1.1 Demographics and Baseline Characteristics

Baseline characteristics will be descriptively summarized for all subjects by treatment group for the ITT population in the Double-blind Segment, and for all subjects in the dose escalation segment by dose. Continuous measures will be summarized with sample size, mean, median, standard deviation, minimum and maximum; categorical measures will be presented with the counts and percents of subjects in each category. No statistical tests comparing treatments at baseline will be performed.

Age is calculated in years after rounding down as follows:

Year of age = (Date informed consent signed - Date of birth) / 365.25

All data will be listed by study segment, treatment group and subject in the double-blind segment and by study segment, dose and subject in the dose escalation segment.

### **10.1.2 Medical History**

Medical history data recorded at screening will be listed by study segment, treatment group and subject in the double-blind segment and by study segment, dose and subject in the dose escalation segment.

# 10.1.3 Inclusion/Exclusion Criteria and Exceptions

Subject inclusion/exclusion criteria and exceptions will be listed by study segment, treatment group and subject in the double-blind segment and by study segment, dose and subject in the dose escalation segment.

#### 10.1.4 Urine Drug Screen

Urine drug screen will be listed by study segment, treatment group and subject in the double-blind segment and by study segment, dose and subject in the dose escalation segment.

#### 10.1.5 Study Drug Administration

Visit, date and time for study drug administration will be listed by study segment, treatment group and subject in the double-blind segment and by study segment, dose and subject in the dose escalation segment.

#### 10.2 Primary Analysis

Efficacy analysis will only be performed for the double-blind randomization segment. FPG from subjects in segment 1 will be presented in by-subject listings.

#### Response Variable and Baseline:

The primary efficacy endpoint of change in FPG will be treated as the response variable. FPG will be determined from the blood samples drawn at baseline, defined as the mean of FPG values on day -2 and day 1 and after 4 weeks of treatment, defined

as the mean of FPG values on day 27 and day 29. If one of the two FPG values at baseline or at 4-week treatment is missing, the single value available will be used. If both values are missing (either baseline or at the 4-week treatment), this data will not be used.

# **Descriptive Summary:**

Descriptive statistics (sample size, mean, median, standard deviation, minimum and maximum) of the primary endpoint will be presented for each treatment group. In addition, descriptive statistics of the baseline and after 4 weeks of treatment values will be presented.

#### ANCOVA Model:

Pairwise comparisons of each active dose versus placebo on mean change in FPG from baseline will be carried out at the two-sided 0.05 alpha level of significance using analysis of covariance adjusting for study center and baseline FPG. Baseline FPG and center will be treated as covariate. The pairwise differences in mean change in FPG means between each dose and placebo, and its associated two-sided 95% confidence interval, adjusted for study center and baseline FPG will be presented.

# **Assessment of Interactions:**

The interactions of treatment-by-baseline and treatment-by-center will be assessed in two separate models using 2 two-way analysis of covariance models with the effects of treatment, center and baseline FPG common to both.

A non-significant interaction effect at the 0.10 level of significance or a significant interaction that is only quantitative and not qualitative in nature (i.e. where the treatment effect differs only in magnitude but not direction across study centers) will support the pooling of subjects across study centers for purposes of the primary analysis pairwise comparisons. Centers with less than 5 subjects randomized will be pooled into one or more centers based on the geographic regions.

#### Missing Data:

No imputation will be carried out for missing data with the exception of subjects who ended treatment due to rescue medication. For such subjects, the last FPG value measured prior to the subject receiving rescue medication will be carried forward to day 29.

#### 10.3 Secondary Analyses

Analysis for the secondary endpoints will be carried out in a similar manner as for the primary efficacy endpoint of FPG. The change in FPG following cessation of treatment will be determined from the blood samples drawn at week 4 of treatment, defined as the mean of FPG values on day 27 and day 29 to week 6, defined as the mean of FPG values on day 41 and day 43. No imputation will be carried out for missing data. Due to the secondary nature of these outcomes, no assessments of the treatment-by-center interaction will be carried out, unless a significant qualitative treatment-by-center interaction is found for FPG. The interaction of treatment-by-baseline, however, will be carried out on all secondary analyses where baseline is measured.

Baseline for weight is defined as the pre-dose weight value on Day 1 at Visit 5. Baseline for HbA1c is defined as the pre-dose HbA1c value on Day 1 at Visit 5. Baseline for 24h UGE is defined as the pre-dose UGE value on Day 0 at Visit 4.

If the safety and ITT analysis sets differ by more than 10%, the analysis on UGE will also be conducted on the safety analysis set.

### 10.4 Safety Analysis

Safety endpoints will be summarized using descriptive statistics and by-subject listings included in the clinical study report. Safety analysis will be performed separately for subjects in the double-blind study and subjects in the dose escalation study where applicable. Results will be presented by treatment group/dose group.

For repeat safety assessments (clinical laboratory tests, vital signs and ECGs), the following will apply for the summary tables.

- Repeat safety assessments prior to dosing, the repeated values will be used for calculations but all values will be included in the listings.
- Repeat safety assessments after dosing, the original values will be used but all values will be included in the listings.

# 10.4.1 Adverse Event Analysis

Adverse events will be mapped using the Medical Dictionary for Regulatory Activities (MedDRA) central coding dictionary (version 12.1). Each adverse event is to be evaluated for date/time of onset, duration, severity and causal relationship with the study drug or other factors.

# **Treatment Emergent Adverse Events**

Treatment Emergent Adverse Events (TEAEs) are any AEs that start or worsen at or after administration of the first dose of study medication.

Adverse Event listings will be provided for all TEAEs, all drug-related TEAEs, serious TEAEs, and any TEAEs leading to study discontinuation.

The number and percentage of subjects experiencing TEAEs will be summarized by treatment group overall and for each System Organ Class and Preferred Term. Each subject will be counted only once within each preferred term. If the same AE occurs in a subject on multiple occasions, the highest severity and least complementary relationship will be assumed. If two or more AEs are reported as a single event, the individual terms will be reported as separate AEs.

This analysis will be repeated for drug-related and serious TEAEs and for TEAEs leading to study discontinuation.

TEAEs will also be tabulated by maximum severity experienced.

No formal statistical tests comparing treatment groups will be performed.

#### Adverse Events during Washout Period

Adverse events reported during the washout period will be presented by subject-listings.

### Serious Adverse Events

Serious adverse events will be listed by-subject listings.

#### Cardiovascular Risk Assessment

Cardiovascular adverse events will be presented in by-subject listings.

### 10.4.2 Clinical Laboratory Tests

Clinical laboratory tests include clinical chemistries, CBC with differential, urinalysis, and urinary electrolytes. These variables will be presented in by-subject listings by study segment, treatment/dose group and subject.

Descriptive statistics (sample size, mean, median standard deviation, minimum, and maximum) of the continuous variables at each visit will be summarized for both double-blind segment and dose escalation segment by treatment/dose group.

Change from baseline to each visit will be presented for double-blind segment. Baseline is defined as the laboratory value prior to dosing. A paired t-test assessing the significance of the change from baseline will be presented for each variable within each treatment group.

Shift tables displaying the change in normality status from baseline to post-baseline visits will be presented for the double-blind segment.

#### 10.4.3 Concomitant Medication

Concomitant medications will be coded using the World Health Organization Dictionary (WHODrug Version 101E). A table of concomitant medications based on the anatomic therapeutic chemical classification (ATC) and preferred name will be produced by treatment/dose group.

A listing of concomitant medications will include all medications taken during the course of the study.

Any medications taken prior to the start of the study medication will be listed and summarized in a similar manner.

No formal statistical tests comparing treatment groups will be performed.

#### 10.4.4 FPG, Vital Signs, SMBG record, and ECG Parameters

Vitals signs including pulse, systolic and diastolic blood pressure at sitting position, respiration rate, and temperature will be measured at screening, prior to dosing, and at each follow up visit.

A 12-lead electrocardiogram (ECG) will be conducted at screening, prior to dosing, and at each follow up visit.

Fasting plasma glucose, vital signs and ECG parameters will be listed and presented in a similar manner as for clinical laboratory tests above.

The SMBG record will be summarized in by-subject listings.

## 10.4.5 Physical Exam

A complete physical examination will be performed at screening and at the termination visit. A complete physical examination will include measurement of body weight and height (height will be measured only at screening), general assessment of all body systems (except genitals) including the skin, head, eyes, ears, nose, throat, neck, thyroid, lungs, heart, abdomen, lymph nodes, and extremities. A partial physical examination will include body weight and general assessment of the skin, heart, lungs and abdomen.

Physical exam will be listed by study segment, treatment group and subject in the doubleblind segment and by study segment, dose and subject in the dose escalation segment.

#### 10.5 PK Assessments

Pharmacokinetic analyses will be performed for EGT0001442 plasma data. All subjects who received EGT0001442 and have sufficient plasma concentration data will be included in the analysis to characterize the PK of EGT0001442. This determination will be made by the study pharmacokineticist.

Subjects who experience emesis will be treated according to Cetero Research SOP entitled "Handling Subjects Experiencing Emesis Episode(s) in BA/BE Studies." Although the SOP's scope is specified as for BA/BE studies, it will be adopted for the analysis of this study, where applicable. Subjects vomiting within 6.6 hours after drug administration will be dropped from the study (based on 2 times the a priori mean population Tmax of 3.3 hours). Their samples will be analyzed by the bioanalytical laboratory and presented in the report but will be excluded from the pharmacokinetic analyses.

Concentration values below the lower limit of quantification (BLQ) will be treated according to Cetero Research SOP entitled "Handling BLQ data in PK/PD studies". Subjects with BLQ values between two non-BLQ concentrations will be set to missing. BLQ values that occur at the beginning on the profile will be set to zero.

Data from subjects with missing concentration values (missed blood draws, lost samples, samples unable to be quantitated) may be used if pharmacokinetic parameters can be estimated using the remaining data points. Otherwise, concentration data from these subjects will be excluded from the final analysis.

A non-compartmental pharmacokinetic analysis (SAS, Cary, NC or WinNonlin 5.0.1, Pharsight Corp., Mountain View, CA, USA) will be used to calculate the PK parameters for each subject. The actual time of sample collection will be used in the PK parameters calculations.

- C<sub>max</sub> Maximum observed plasma concentration
- T<sub>max</sub> Time of observed maximum plasma concentration
- Kel Terminal phase rate constant
- Thalf Apparent terminal half life
- CL/F The apparent total body clearance

- V<sub>7</sub>/F The apparent total volume of distribution
- AUC<sub>0-t</sub> Area under the plasma concentration-time curve from Time 0 to Time t (time of last quantifiable plasma concentration)
- AUC<sub>0-inf</sub> Area under the plasma concentration-time curve from Time 0 to infinity
- AUC<sub>0-24</sub> Area under the plasma concentration-time curve from Time 0 to 24 h

Descriptive statistics (arithmetic mean, standard deviation [sd], median, minimum, maximum, coefficient of variation) will be summarized by dose group for the parameters listed above and for In-AUC $_{0-t}$ , In-AUC $_{0-24}$ , In-AUC $_{0-inf}$  and In-C $_{max}$ . Additionally, geometric means will be calculated for AUC $_{0-t}$ , AUC $_{0-24}$ , AUC $_{0-inf}$  and C $_{max}$ .

No value of Kel,  $AUC_{0-inf}$ , Thalf, CL/F, or  $V_z/F$  will be reported for cases that do not exhibit a terminal log-linear phase in the concentration versus time profile.

Other pharmacokinetic parameters may be calculated if deemed necessary.

### 10.6 Exploratory Analysis of the Post-prandial Blood Glucose

The impact of EGT0001442 on 2-h post-prandial glucose levels will be determined by measuring fingerstick blood glucose values at 7 points on day 0 and then again on day 2 of drug administration for the 20 subjects in the dose escalation phase of the trial. Measurements will be taken before each meal (breakfast, lunch, and dinner) and then 2 hour after meal completion. A seventh measurement will be taken at 10 pm ( $\pm$  30 mins) at night.

The difference between the post-meal measurement and the measurement before the same meal will be identified as the post-prandial glucose change for that meal. For each meal, the difference in day 0 to day 2 post-prandial glucose changes will be descriptively summarized for all subjects in the dose escalation segment, categorized by dose. The data will be summarized with sample size, mean, median, standard deviation, minimum and maximum. No statistical tests comparing doses will be performed

For each subject, AUC of the glucose levels across the 7 points will be calculated at each of day 0 and day 2. The difference in day 0 to day 2 AUC will be descriptively summarized for all subjects in the dose escalation segment, categorized by dose. The data will be summarized with sample size, mean, median, standard deviation, minimum and maximum. No statistical tests comparing doses will be performed.

# 10.7 Interim Analysis

There will be no formal interim efficacy analysis for this study. An independent data and safety monitoring board (DSMB) will inspect the safety data from the dose escalation segment, review SAE reports, and will periodically inspect unblinded safety data from the double-blind study. A DSMB charter will be written outlining the safety data to be inspected periodically by the DSMB.

## 10.8 Missing Data

No imputation will be carried out for missing data with the exception of subjects who ended treatment due to rescue medication. For such subjects, the last FPG value measured prior to the subject receiving rescue medication will be carried forward to Day 28.

# 10.9 Multiple Comparisons

Given the Phase II nature of this study, no adjustment of the significance level for multiple comparisons will be made.

#### 11. TABLE, LISTING AND FIGURE SHELLS

The following shells are provided in order to provide a framework for the display of data from this study. The shells may change due to unforeseen circumstances. These shells may not be reflective of every aspect of this study but are intended to show the general layout of the Tables, Listings and Figures that will be included in the final report. Tables and listings are numbered following the ICH structure. Table headers, variables names and footnotes will be modified as needed following data analyses. Please note that all summary tables and listings will be generated using SAS® Version 9.1.3. Figures will be generated using SigmaPlot Version 10 and/or SAS® Version 9.1.3.

# **Summary Tables**

Table 14.1.1 Disposition of Subjects (Double-blind Segment)

| | | | Treatmen | t Group | | |
|---|---|---|---|---|---|---|
| | Placebo<br>(N=xx) | EGT0001442<br>5 mg<br>(N=xx) | EGT0001442<br>10 mg<br>(N=xx) | EGT0001442<br>20 mg<br>(N=xx) | EGT0001442<br>50 mg<br>(N=xx) | Overall<br>(N=xx) |
| Number of subjects randomized (N) | XX | xx | XX | XX | XX | XX |
| <pre>Included in Double-blind Safety Analysis Set [n (%)]</pre> | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) |
| <pre>Included in Intent-to-Treat Analysis Set [n (%)]</pre> | xx (xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) |
| Included in Per-Protocol Analysis Set [n (%)] | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) |
| <pre>Included in Completed study [n (%)]</pre> | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) |
| Discontinued from study [n (%)] | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) |
| Reason for Discontinuation | | | | | | |
| Discontinued due to Adverse Event [n (%)] | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) |
| Subject elected to withdraw from study [n (%)] | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) |
| Death [n (%)] | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) |
| Study terminated by sponsor [n (%)] | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) |
| <pre>Investigator decision [n (%)]</pre> | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) |
| Lost to follow-up [n (%)] | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) |
| Poor Glycemic Control [n (%)] | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) |
| Other [n (%)] | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) |

N: Number of subjects randomized in the specified treatment group

n: Number of subjects

<sup>%:</sup> Percentage based on N

Table 14.1.2 Disposition of Subjects (Dose Escalation Segment)

| | Dose Group | | | | |
|---|---|---|---|---|---|
| | EGT0001442<br>5 mg<br>(N=xx) | EGT0001442<br>10 mg<br>(N=xx) | EGT0001442<br>20 mg<br>(N=xx) | EGT0001442<br>50 mg<br>(N=xx) | Overall (N=xx) |
| Number of subjects enrolled (N) | XX | XX | xx | XX | xx |
| Included in Dose-Escalation Safety Analysis Set [n ( | %)] xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) |
| Included in Completed study [n (%)] | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x% |
| Discontinued from study [n (%)] | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x% |
| Reason for Discontinuation | | | | | |
| Discontinued due to Adverse Event [n (%)] | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) |
| Subject elected to withdraw from study [n (%)] | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) |
| Death [n (%)] | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) |
| Study terminated by sponsor [n (%)] | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x% |
| <pre>Investigator decision [n (%)]</pre> | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) |
| Lost to follow-up [n (%)] | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) |
| Other [n (%)] | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) |

N: Number of subjects enrolled in the specified dose group

n: Number of subjects

<sup>%:</sup> Percentage based on N

Table 14.1.3 Summary of Demographics (Double-blind Segment)

| Parameter | Statistic | Placebo<br>(N=xx) | EGT0001442<br>5 mg<br>(N=xx) | EGT0001442<br>10 mg<br>(N=xx) | EGT0001442<br>20 mg<br>(N=xx) | EGT0001442<br>50 mg<br>(N=xx) | Overall (N=xx) |
|---|---|---|---|---|---|---|---|
| Age (years) | n | XX | XX | xx | xx | XX | XX |
| | Mean ± SD | $xx \pm x.x$ | $xx \pm x.x$ | xx ± x.x | $xx \pm x.x$ | $xx \pm x.x$ | $xx \pm x.x$ |
| | Median | XX | XX | XX | XX | XX | XX |
| | Min , Max | xx , xx | xx , xx | xx , xx | xx , xx | xx , xx | xx , xx |
| Height (cm) | n | XX | xx | xx | xx | XX | xx |
| _ | Mean ± SD | $xx.x \pm x.xx$ | $xx.x \pm x.xx$ | $xx.x \pm x.xx$ | $xx.x \pm x.xx$ | $xx.x \pm x.xx$ | $xx.x \pm x.xx$ |
| | Median | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| | Min , Max | xx.x , xx.x | xx.x , xx.x | xx.x , xx.x | xx.x , xx.x | xx.x , xx.x | xx.x , xx.x |
| Weight (kg) | n | XX | XX | XX | XX | XX | XX |
| 3 . 3. | Mean ± SD | $xx.x \pm x.xx$ | xx.x ± x.xx | xx.x ± x.xx | $xx.x \pm x.xx$ | $xx.x \pm x.xx$ | $xx.x \pm x.xx$ |
| | Median | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| | Min , Max | XX.X , XX.X | xx.x , xx.x | xx.x , xx.x | xx.x , xx.x | xx.x , xx.x | xx.x , xx.x |
| BMI (kg/m^2) | n | XX | XX | XX | XX | XX | XX |
| , | Mean ± SD | $xx.x \pm x.xx$ | xx.x ± x.xx | xx.x ± x.xx | $xx.x \pm x.xx$ | xx.x ± x.xx | $xx.x \pm x.xx$ |
| | Median | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| | Min , Max | XX.X , XX.X | xx.x , xx.x | XX.X , XX.X | xx.x , xx.x | xx.x , xx.x | xx.x , xx.x |

N: Number of subjects randomized in the specified treatment group

n: Number of subjects

SD: Standard Deviation

Table 14.1.3 Summary of Demographics (Double-blind Segment) (continued)

Treatment Group EGT0001442 EGT0001442 EGT0001442 EGT0001442 Placebo 5 mg 20 mg 50 mg Overall 10 mg Statistic (N=xx)(N=xx)(N=xx)(N=xx)Parameter (N=xx)(N=xx)Race [n (%)] American Indian / Alaska Native xx(xx.x%) xx(xx.x%) xx(xx.x%) xx(xx.x%) xx(xx.x%) xx(xx.x%) Asian xx(xx.x%) xx(xx.x%) xx(xx.x%) xx(xx.x%) xx(xx.x%) xx(xx.x%) Black / African American xx(xx.x%) xx(xx.x%) xx(xx.x%) xx(xx.x%) xx(xx.x%) xx(xx.x%) Native Hawaiian / Other Pacific Islander xx(xx.x%) xx(xx.x%) xx(xx.x%) xx(xx.x%) xx(xx.x%) xx(xx.x%) White xx(xx.x%) xx(xx.x%) xx(xx.x%) xx(xx.x%) xx(xx.x%) xx(xx.x%) Gender [n (%)] Male xx(xx.x%) xx(xx.x%) xx(xx.x%) xx(xx.x%) xx(xx.x%) xx(xx.x%) Female xx(xx.x%) xx(xx.x%) xx(xx.x%) xx(xx.x%) xx(xx.x%) xx(xx.x%) Ethnicity [n (%)] Hispanic or Latino xx(xx.x%) xx(xx.x%) xx(xx.x%) xx(xx.x%) xx(xx.x%) xx(xx.x%) Not Hispanic or Latino xx(xx.x%) xx(xx.x%) xx(xx.x%) xx(xx.x%) xx(xx.x%) xx(xx.x%)

N: Number of subjects randomized in the specified treatment group

n: Number of subjects

<sup>%:</sup> Percentage based on N

Table 14.1.4 Summary of Demographics (Dose Escalation Segment)

Treatment Group EGT0001442 EGT0001442 EGT0001442 EGT0001442 5 mg 10 mg 20 mg 50 mg Overall Statistic (N=xx)(N=xx)(N=xx)Parameter (N=xx)(N=xx)Age (years) XX XX XX XX Mean ± SD xx ± x.x xx ± x.x xx ± x.x xx ± x.x  $xx \pm x.x$ Median XX XX XX XX XX Min , Max XX , XX XX , XX XX , XX XX , XX XX , XX Height (cm) XX XX XX XX Mean ± SD  $xx.x \pm x.xx$ xx.x ± x.xx  $xx.x \pm x.xx$  $xx.x \pm x.xx$ xx.x ± x.xx Median XX.X XX.X XX.X XX.X XX.X Min , Max XX.X , XX.X XX.X , XX.X XX.X , XX.X XX.X , XX.X xx.x , xx.x Weight (kg) XX XX Mean ± SD xx.x ± x.xx  $xx.x \pm x.xx$  $xx.x \pm x.xx$  $xx.x \pm x.xx$  $xx.x \pm x.xx$ Median XX.X XX.X XX.X XX.X XX.X Min , Max xx.x , xx.x XX.X , XX.X XX.X , XX.X xx.x , xx.x xx.x , xx.x BMI  $(kq/m^2)$ Mean ± SD xx.x ± x.xx  $xx.x \pm x.xx$  $xx.x \pm x.xx$  $xx.x \pm x.xx$ xx.x ± x.xx

XX.X

XX.X , XX.X XX.X , XX.X XX.X , XX.X

XX.X

XX.X

XX.X

XX.X , XX.X XX.X , XX.X

XX.X

Median

Min , Max

N: Number of subjects enrolled in the specified dose group

n: Number of subjects SD: Standard Deviation

<sup>(</sup>Source: path\program name Date/time of run: ddmmmyyyy:hh:mm)

Table 14.1.4 Summary of Demographics (Dose Escalation Segment) (continued)

| Parameter | | Treatment Group | | | | |
|---|---|---|---|---|---|---|
| | Statistic | EGT0001442<br>5 mg<br>(N=xx) | EGT0001442<br>10 mg<br>(N=xx) | EGT0001442<br>20 mg<br>(N=xx) | EGT0001442<br>50 mg<br>(N=xx) | Overall (N=xx) |
| Race | [n (%)] | | | | | |
| American Indian | / Alaska Native | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) |
| Asian | | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) |
| Black / African . | American | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) |
| Native Hawaiian | / Other Pacific Islander | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) |
| White | | xx (xx.x%) | xx(xx.x%) | xx (xx.x%) | xx (xx.x%) | xx(xx.x%) |
| ender | [n (%)] | | | | | |
| Male | | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) |
| Female | | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) |
| Sthnicity | [n (%)] | | | | | |
| Hispanic or Lati | no | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) |
| Not Hispanic or | Latino | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) |

N: Number of subjects randomized in the specified treatment group

n: Number of subjects

<sup>%:</sup> Percentage based on N

Table 14.2.1 Primary Efficacy Analysis: Descriptive Summary of Fasting Plasma Glucose from Baseline to End of Treatment
Double-blind Segment
Intent-to-Treat Analysis Set

| | | Treatment Group | | | | |
|---|---|---|---|---|---|---|
| | Statistic | Placebo<br>(N=xx) | EGT0001442<br>5 mg<br>(N=xx) | EGT0001442<br>10 mg<br>(N=xx) | EGT0001442<br>20 mg<br>(N=xx) | EGT0001442<br>50 mg<br>(N=xx) |
| Baseline* | n | xx | xx | xx | xx | xx |
| | Mean ± SD | $xx.x \pm x.xx$ | $xx.x \pm x.xx$ | $xx.x \pm x.xx$ | $xx.x \pm x.xx$ | $xx.x \pm x.xx$ |
| | Median | XX.X | xx.x | xx.x | XX.X | XX.X |
| | Min, Max | xx , xx | xx , xx | xx , xx | xx , xx | xx , xx |
| End of Treatment# | n | xx | XX | xx | xx | xx |
| | Mean ± SD | $xx.x \pm x.xx$ | $xx.x \pm x.xx$ | $xx.x \pm x.xx$ | $xx.x \pm x.xx$ | $xx.x \pm x.xx$ |
| | Median | XX.X | XX.X | XX.X | XX.X | XX.X |
| | Min, Max | xx , xx | XX , XX | xx , xx | xx , xx | xx , xx |
| Change from Baseline to | n | xx | XX | xx | xx | xx |
| End of Treatment | Mean ± SD | $xx.x \pm x.xx$ | $xx.x \pm x.xx$ | $xx.x \pm x.xx$ | $xx.x \pm x.xx$ | $xx.x \pm x.xx$ |
| | Median | XX.X | XX.X | XX.X | XX.X | XX.X |
| | Min, Max | xx , xx | xx , xx | xx , xx | xx , xx | xx , xx |

Note: \* Baseline is defined as the mean of FPG values on day -2 and day 1.

<sup>#</sup> End of Treatment is defined as the mean of FPG values on day 27 and day 29.

Table 14.2.2 Primary Efficacy Analysis: ANCOVA Results on Mean Change in FPG from Baseline to End of Treatment

Double-blind Segment

Intent-to-Treat Analysis Set

| Treatment | n | LSMeans | Std Err<br>LSMeans | LSMeans | Std Err<br>LSMeans | 95%-confidence<br>Interval | P-value<br>Treatment | P-value<br>Baseline | P-value<br>Center |
|---|---|---|---|---|---|---|---|---|---|
| Overall | xxx | | | | | | x.xxxx | x.xxxx | x.xxxx |
| Placebo | XXX | x.xxx | x.xxx | | | | | | |
| 5 mg EGT0001442 vs. Placebo | XXX | x.xxx | x.xxx | x.xxx | x.xxx | x.xxx, x.xxx | x.xxxx | | |
| 10 mg EGT0001442 vs. Placebo | XXX | x.xxx | x.xxx | x.xxx | x.xxx | x.xxx, x.xxx | x.xxxx | | |
| 20 mg EGT0001442 vs. Placebo | XXX | x.xxx | x.xxx | x.xxx | x.xxx | x.xxx, x.xxx | x.xxxx | | |
| 50 mg EGT0001442 vs. Placebo | XXX | x.xxx | x.xxx | x.xxx | x.xxx | x.xxx, x.xxx | x.xxxx | | |

n: Number of subjects with data available in the specific treatment group

LSMeans: Least square means

Std Err LSMeans: Standard error of the LSMeans

Note: LSMeans, Std Err of LSMeans, 95% confidence intervals and p-values are based on an ANCOVA with change from baseline as

dependent variable and treatment as fixed effect and baseline and center as covariates. P-values are from two-sided test

at 5%-level.

Note: Baseline is defined as the mean of FPG values on day -2 and day 1.

End of Treatment is defined as the mean of FPG values on day 27 and day 29.

# Similar tables:

Table 14.2.3 Descriptive Summary of Fasting Plasma Glucose from Baseline to End of Treatment
Double-blind Segment
Per-Protocol Analysis Set

Table 14.2.4 ANCOVA Results on Mean Change in FPG from Baseline to End of Treatment
Double-blind Segment
Per-Protocol Analysis Set

Table 14.2.5 Descriptive Summary of Fasting Plasma Glucose from End of Treatment to Post Treatment

Double-blind Segment

Intent-to-Treat Analysis Set

| | | Treatment Group | | | | |
|---|---|---|---|---|---|---|
| | Statistic | Placebo<br>(N=xx) | EGT0001442<br>5 mg<br>(N=xx) | EGT0001442<br>10 mg<br>(N=xx) | EGT0001442<br>20 mg<br>(N=xx) | EGT0001442<br>50 mg<br>(N=xx) |
| End of Treatment# | n | xx | xx | xx | xx | XX |
| | Mean ± SD | $xx.x \pm x.xx$ | $xx.x \pm x.xx$ | $xx.x \pm x.xx$ | $xx.x \pm x.xx$ | $xx.x \pm x.xx$ |
| | Median | XX.X | XX.X | XX.X | XX.X | XX.X |
| | Min, Max | XX , XX | xx , xx | XX , XX | XX , XX | xx , xx |
| Post Treatment+ | n | xx | XX | XX | XX | xx |
| | Mean ± SD | $xx.x \pm x.xx$ | $xx.x \pm x.xx$ | $xx.x \pm x.xx$ | $xx.x \pm x.xx$ | $xx.x \pm x.xx$ |
| | Median | XX.X | XX.X | XX.X | XX.X | XX.X |
| | Min, Max | xx , xx | xx , xx | xx , xx | xx , xx | xx , xx |
| Change from End of Treatment to | n | xx | XX | xx | xx | xx |
| Post Treatment | Mean ± SD | $xx.x \pm x.xx$ | $xx.x \pm x.xx$ | $xx.x \pm x.xx$ | $xx.x \pm x.xx$ | $xx.x \pm x.xx$ |
| | Median | XX.X | XX.X | XX.X | XX.X | XX.X |
| | Min, Max | XX , XX | XX , XX | XX , XX | xx , xx | XX , XX |

Note: # End of Treatment is defined as the mean of FPG values on day 27 and day 29.

<sup>+</sup> Post Treatment is determined from the blood samples drawn at week 4 of treatment, defined as the mean of FPG values on day 27 and day 29 to week 6, defined as the mean of FPG values on day 41 and day 43.

# Table 14.2.6 ANCOVA Results on Mean Change in FPG from End of Treatment to Post Treatment Double-blind Segment Intent-to-Treat Analysis Set

| Treatment | n | LSMeans | Std Err<br>LSMeans | LSMeans | Std Err<br>LSMeans | 95%-confidence<br>Interval | P-value<br>Treatment | P-value<br>Baseline | P-value<br>Center |
|---|---|---|---|---|---|---|---|---|---|
| Overall | xxx | | | | | | x.xxxx | x.xxxx | x.xxxx |
| Placebo | xxx | x.xxx | x.xxx | | | | | | |
| 5 mg EGT0001442 vs. Placebo | xxx | x.xxx | x.xxx | x.xxx | x.xxx | x.xxx, x.xxx | x.xxxx | | |
| 10 mg EGT0001442 vs. Placebo | xxx | x.xxx | x.xxx | x.xxx | x.xxx | x.xxx, x.xxx | x.xxxx | | |
| 20 mg EGT0001442 vs. Placebo | xxx | x.xxx | x.xxx | x.xxx | x.xxx | x.xxx, x.xxx | x.xxxx | | |
| 50 mg EGT0001442 vs. Placebo | xxx | x.xxx | x.xxx | x.xxx | x.xxx | x.xxx, x.xxx | x.xxxx | | |

n: Number of subjects with data available in the specific treatment group

LSMeans: Least square means

Std Err LSMeans: Standard error of the LSMeans

Note: LSMeans, Std Err of LSMeans, 95% confidence intervals and p-values are based on an ANCOVA with change from baseline as dependent variable and treatment as fixed effect and baseline and center as covariates. P-values are from two-sided test

at 5%-level. Note: End of Treatment is defined as the mean of FPG values on day 27 and day 29.

Post Treatment is determined from the blood samples drawn at week 4 of treatment, defined as the mean of FPG values on day 27 and day 29 to week 6, defined as the mean of FPG values on day 41 and day 43.

Table 14.2.7 Descriptive Summary of Change in Body Weight from Baseline to Day 29

Double-blind Segment

Intent-to-Treat Analysis Set

| | Statistic | | Treatment Group | | | |
|---|---|---|---|---|---|---|
| | | Placebo<br>(N=xx) | EGT0001442<br>5 mg<br>(N=xx) | EGT0001442<br>10 mg<br>(N=xx) | EGT0001442<br>20 mg<br>(N=xx) | EGT0001442<br>50 mg<br>(N=xx) |
| Baseline | n | xx | xx | xx | xx | xx |
| | Mean ± SD | xx.x ± x.xx | xx.x ± x.xx | xx.x ± x.xx | xx.x ± x.xx | xx.x ± x.xx |
| | Median | xx.x | xx.x | xx.x | xx.x | xx.x |
| | Min, Max | XX , XX | xx , xx | xx , xx | xx , xx | xx , xx |
| Day 29 | n | xx | xx | xx | xx | xx |
| | Mean ± SD | xx.x ± x.xx | xx.x ± x.xx | xx.x ± x.xx | xx.x ± x.xx | xx.x ± x.xx |
| | Median | xx.x | xx.x | xx.x | xx.x | xx.x |
| | Min, Max | xx , xx | xx , xx | xx , xx | xx , xx | xx , xx |
| Change from baseline | n | xx | xx | xx | xx | xx |
| | Mean ± SD | xx.x ± x.xx | xx.x ± x.xx | xx.x ± x.xx | xx.x ± x.xx | xx.x ± x.xx |
| | Median | xx.x | xx.x | xx.x | xx.x | xx.x |
| | Min, Max | xx , xx | xx , xx | xx , xx | xx , xx | xx , xx |

Note: Baseline is defined as the pre-dose body weight value on Day 1.

# Table 14.2.8 ANCOVA Results on Mean Change in Body Weight from Baseline to Day 29 Double-blind Segment Intent-to-Treat Analysis Set

| | | Difference between Treatments | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|
| Treatment | n | LSMeans | Std Err<br>LSMeans | LSMeans | Std Err<br>LSMeans | 95%-confidence<br>Interval | P-value<br>Treatment | P-value<br>Baseline | P-value<br>Center |
| Overall | xxx | | | | | | x.xxx | x.xxx | x.xxxx |
| Placebo | xxx | x.xxx | x.xxx | | | | | | |
| 5 mg EGT0001442 vs. Placebo | xxx | x.xxx | x.xxx | x.xxx | x.xxx | x.xxx, x.xxx | x.xxxx | | |
| 10 mg EGT0001442 vs. Placebo | xxx | x.xxx | x.xxx | x.xxx | x.xxx | x.xxx, x.xxx | x.xxxx | | |
| 20 mg EGT0001442 vs. Placebo | xxx | x.xxx | x.xxx | x.xxx | x.xxx | x.xxx, x.xxx | x.xxxx | | |
| 50 mg EGT0001442 vs. Placebo | XXX | x.xxx | x.xxx | x.xxx | x.xxx | x.xxx, x.xxx | x.xxxx | | |

n: Number of subjects with data available in the specific treatment group

LSMeans: Least square means

Std Err LSMeans: Standard error of the LSMeans

Note: LSMeans, Std Err of LSMeans, 95% confidence intervals and p-values are based on an ANCOVA with change from baseline as dependent variable and treatment as fixed effect and baseline and center as covariates. P-values are from two-sided test

at 5%-level.

Note: Baseline is defined as the pre-dose body weight value on Day 1.

Table 14.2.9 Descriptive Summary of Change in HbA1c from Baseline to Day 29

Double-blind Segment

Intent-to-Treat Analysis Set

| | Statistic | Treatment Group | | | | |
|---|---|---|---|---|---|---|
| | | Placebo<br>(N=xx) | EGT0001442<br>5 mg<br>(N=xx) | EGT0001442<br>10 mg<br>(N=xx) | EGT0001442<br>20 mg<br>(N=xx) | EGT0001442<br>50 mg<br>(N=xx) |
| Baseline | n<br>Mean ± SD<br>Median | xx<br>xx.x ± x.xx | xx<br>xx.x ± x.xx | xx<br>xx.x ± x.xx | xx<br>xx.x ± x.xx | xx<br>xx.x ± x.xx |
| | Median<br>Min, Max | xx.x<br>xx , xx | xx.x<br>xx , xx | xx.x<br>xx, xx | xx.x<br>xx , xx | xx.x<br>xx, xx |
| Day 29 | n<br>Mean ± SD<br>Median<br>Min, Max | xx<br>xx.x ± x.xx<br>xx.x<br>xx , xx | xx<br>xx.x ± x.xx<br>xx.x<br>xx , xx | xx<br>xx.x ± x.xx<br>xx.x<br>xx , xx | xx<br>xx.x ± x.xx<br>xx.x<br>xx , xx | xx<br>xx.x ± x.xx<br>xx.x<br>xx , xx |
| Change from baseline | n<br>Mean ± SD<br>Median<br>Min, Max | xx<br>xx.x ± x.xx<br>xx.x<br>xx , xx | xx<br>xx.x ± x.xx<br>xx.x<br>xx , xx | xx<br>xx.x ± x.xx<br>xx.x<br>xx , xx | xx<br>xx.x ± x.xx<br>xx.x<br>xx , xx | xx<br>xx.x ± x.xx<br>xx.x<br>xx , xx |

Note: Baseline is defined as the pre-dose HbAlc value on Day 1.
### Table 14.2.10 ANCOVA Results on Mean Change in HbA1c from Baseline to Day 29 Double-blind Segment Intent-to-Treat Analysis Set

| | | | | | Difference | e between Treatme | nts | | |
|---|---|---|---|---|---|---|---|---|---|
| Treatment | n | LSMeans | Std Err<br>LSMeans | LSMeans | Std Err<br>LSMeans | 95%-confidence<br>Interval | P-value<br>Treatment | P-value<br>Baseline | P-value<br>Center |
| Overall | xxx | | | | | | x.xxxx | x.xxxx | x.xxx |
| Placebo | xxx | x.xxx | x.xxx | | | | | | |
| 5 mg EGT0001442 vs. Placebo | XXX | x.xxx | x.xxx | x.xxx | x.xxx | x.xxx, x.xxx | x.xxxx | | |
| 10 mg EGT0001442 vs. Placebo | xxx | x.xxx | x.xxx | x.xxx | x.xxx | x.xxx, x.xxx | x.xxxx | | |
| 20 mg EGT0001442 vs. Placebo | xxx | x.xxx | x.xxx | x.xxx | x.xxx | x.xxx, x.xxx | x.xxxx | | |
| 50 mg EGT0001442 vs. Placebo | XXX | x.xxx | x.xxx | x.xxx | x.xxx | x.xxx, x.xxx | x.xxxx | | |

n: Number of subjects with data available in the specific treatment group

LSMeans: Least square means

Std Err LSMeans: Standard error of the LSMeans

Note: LSMeans, Std Err of LSMeans, 95% confidence intervals and p-values are based on an ANCOVA with change from baseline as

dependent variable and treatment as fixed effect and baseline and center as covariates. P-values are from two-sided test

at 5%-level.

Note: Baseline is defined as the pre-dose HbAlc value on Day 1.

Table 14.2.11 Descriptive Summary of Change in 24 h UGE from Baseline to Day 28

Double-blind Segment

Intent-to-Treat Analysis Set

| | | | | Treatment Group | | |
|---|---|---|---|---|---|---|
| | Statistic | Placebo<br>(N=xx) | EGT0001442<br>5 mg<br>(N=xx) | EGT0001442<br>10 mg<br>(N=xx) | EGT0001442<br>20 mg<br>(N=xx) | EGT0001442<br>50 mg<br>(N=xx) |
| Baseline | n<br>Mean ± SD<br>Median<br>Min, Max | xx<br>xx.x ± x.xx<br>xx.x<br>xx , xx | xx<br>xx.x ± x.xx<br>xx.x<br>xx , xx | xx<br>xx.x ± x.xx<br>xx.x<br>xx , xx | xx<br>xx.x ± x.xx<br>xx.x<br>xx , xx | xx<br>xx.x ± x.xx<br>xx.x<br>xx , xx |
| Day 1 | n<br>Mean ± SD<br>Median<br>Min, Max | xx<br>xx.x ± x.xx<br>xx.x<br>xx , xx | xx<br>xx.x ± x.xx<br>xx.x<br>xx , xx | xx<br>xx.x ± x.xx<br>xx.x<br>xx , xx | xx<br>xx.x ± x.xx<br>xx.x<br>xx , xx | xx<br>xx.x ± x.xx<br>xx.x<br>xx , xx |
| Day 28 | n<br>Mean ± SD<br>Median<br>Min, Max | xx<br>xx.x ± x.xx<br>xx.x<br>xx , xx | xx<br>xx.x ± x.xx<br>xx.x<br>xx , xx | xx<br>xx.x ± x.xx<br>xx.x<br>xx , xx | xx<br>xx.x ± x.xx<br>xx.x<br>xx , xx | xx<br>xx.x ± x.xx<br>xx.x<br>xx , xx |
| Change from baseline<br>to Day 1 | n<br>Mean ± SD<br>Median<br>Min, Max | xx<br>xx.x ± x.xx<br>xx.x<br>xx , xx | xx<br>xx.x ± x.xx<br>xx.x<br>xx , xx | xx<br>xx.x ± x.xx<br>xx.x<br>xx , xx | xx<br>xx.x ± x.xx<br>xx.x<br>xx , xx | xx<br>xx.x ± x.xx<br>xx.x<br>xx , xx |
| Change from baseline<br>to Day 28 | n<br>Mean ± SD<br>Median<br>Min, Max | xx<br>xx.x ± x.xx<br>xx.x<br>xx , xx | xx<br>xx.x ± x.xx<br>xx.x<br>xx , xx | xx<br>xx.x ± x.xx<br>xx.x<br>xx , xx | xx<br>xx.x ± x.xx<br>xx.x<br>xx , xx | xx<br>xx.x ± x.xx<br>xx.x<br>xx , xx |

Note: Baseline is defined as the 24h UGE on Day 0.

### Table 14.2.12 ANCOVA Results on Mean Change in 24 h UGE from Baseline to Day 28 Double-blind Segment Intent-to-Treat Analysis Set

| | | | | | Difference | e between Treatme | nts | | |
|---|---|---|---|---|---|---|---|---|---|
| Treatment | n | LSMeans | Std Err<br>LSMeans | LSMeans | Std Err<br>LSMeans | 95%-confidence<br>Interval | P-value<br>Treatment | P-value<br>Baseline | P-value<br>Center |
| Overall | xxx | | | | | | x.xxxx | x.xxxx | x.xxxx |
| Placebo | XXX | x.xxx | x.xxx | | | | | | |
| 5 mg EGT0001442 vs. Placebo | XXX | x.xxx | x.xxx | x.xxx | x.xxx | x.xxx, x.xxx | x.xxxx | | |
| 10 mg EGT0001442 vs. Placebo | XXX | x.xxx | x.xxx | x.xxx | x.xxx | x.xxx, x.xxx | x.xxxx | | |
| 20 mg EGT0001442 vs. Placebo | XXX | x.xxx | x.xxx | x.xxx | x.xxx | x.xxx, x.xxx | x.xxxx | | |
| 50 mg EGT0001442 vs. Placebo | XXX | x.xxx | x.xxx | X.XXX | x.xxx | x.xxx, x.xxx | x.xxxx | | |

n: Number of subjects with data available in the specific treatment group

LSMeans: Least square means

Std Err LSMeans: Standard error of the LSMeans

Note: LSMeans, Std Err of LSMeans, 95% confidence intervals and p-values are based on an ANCOVA with change from baseline as

dependent variable and treatment as fixed effect and baseline and center as covariates. P-values are from two-sided test

at 5%-level.

Note: Baseline is defined as the 24h UGE on Day 0.

Table 14.2.13 Summary of Plasma Concentrations of EGT0001442 (ng/mL)

Dose Escalation Segment

| Dose | | Subject | 0 | 0.5 | 1 | 2 | 3 | 4 | 6 | 8 | 10 | 12 | 24 | 48 |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Group | Center | Number | hr | hr | hr | hr | hr | hr | hr | hr | hr | hr | hr | hr |
| 5 mg EGT0001442 | 01 | 01 | XXXX | XXXX | XXXX | XXXX | XXXX | XXXX | XXXX | XXXX | XXXX | XXXX | XXXX | XXXX |
| | | 02 | XXXX | XXXX | XXXX | XXXX | XXXX | XXXX | XXXX | XXXX | XXXX | XXXX | XXXX | XXXX |
| | | 03 | XXXX | XXXX | XXXX | XXXX | XXXX | XXXX | XXXX | XXXX | XXXX | XXXX | XXXX | XXXX |
| | | N | xx | XX | XX | XX | xx | xx | XX | XX | XX | XX | XX | XX |
| | | MEAN | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| | | SD | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| | | CV% | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| | | MEDIAN | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| | | MIN | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| | | MAX | XX.XX | XX.XX | xx.xx | XX.XX | xx.xx | xx.xx | XX.XX | xx.xx | xx.xx | XX.XX | xx.xx | XX.XX |

Note: table will continue for 10mg, 20mg and 50mg dose groups.

Table 14.2.14 Summary of Pharmacokinetic Parameters of EGT0001442

Dose Escalation Segment

| | | | | | | | | | | | | Ln-Transf | ormed | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Dose | Subject | AUC0-t | AUC0-24 | AUC0-inf | Cmax | Tmax | Thalf | Kel | Vz/F | CL/F | AUC0-t | AUC0-24 | AUC0-inf | Cmax |
| Group | Number | (ng.h/mL) | (ng.h/mL) | (ng.h/mL) | (ng/mL) | (h) | (h) | (1/h) | (L) | (L/h) | (ng.h/mL | ) (ng.h/mL) | (ng.h/mL) | (ng/mL) |
| 5 mg EGT0001442 | 01 | XXXX.X | XXXX.X | XXXX.X | XXX.X | XX.X | XX.X | x.xx | XX | xxx.x | XXX.X | XXX.X | XXX.X | XXX.X |
| | 02 | XXXX.X | XXXX.X | XXXX.X | XXX.X | XX.X | XX.X | X.XX | XX | xxx.x | XXX.X | XXX.X | XXX.X | xxx.x |
| 1 | 1 | xxxx.x | xxxx.x | xxxx.x | xxx.x | XX.X | XX.X | x.xx | XX : | xxx.x | xxx.x | xxx.x | xxx.x | XXX.X |
| I | 1EAN | XXXX.X | xxxx.x | XXXX.X | xxx.x | XX.X | XX.X | X.XX | XX : | XXX.X | xxx.x | XXX.X | XXX.X | XXX.X |
| S | SD | XXXX.X | XXXX.X | XXXX.X | XXX.X | XX.X | XX.X | X.XX | XX : | XXX.X | XXX.X | XXX.X | XXX.X | XXX.X |
| ( | CV% | XXXX.X | xxxx.x | XXXX.X | xxx.x | XX.X | XX.X | X.XX | XX : | XXX.X | xxx.x | XXX.X | XXX.X | XXX.X |
| I | MEDIAN | XXXX.X | xxxx.x | XXXX.X | xxx.x | XX.X | XX.X | X.XX | XX : | XXX.X | xxx.x | XXX.X | XXX.X | XXX.X |
| I | MIN | xxxx.x | xxxx.x | xxxx.x | XXX.X | XX.X | XX.X | X.XX | XX : | xxx.x | xxx.x | XXX.X | XXX.X | XXX.X |
| I | IAX | XXXX.X | xxxx.x | XXXX.X | xxx.x | XX.X | XX.X | X.XX | XX : | XXX.X | xxx.x | XXX.X | XXX.X | XXX.X |
| ( | SM* | xxxx.x | xxxx.x | XXXX.X | xxx.x | | | | | | | | | |

Note: \*GM = Geometric Mean

Note: table will continue for 10mg, 20mg and 50mg dose groups.

Table 14.2.15 Summary of Post Prandial Blood Glucose (mg/dL) in Change from Day 0 to Day 2

Dose Escalation Segment

| | | | | Dose Group | | |
|---|---|---|---|---|---|---|
| Day | Meal | -<br>Statistic | EGT0001442<br>5 mg<br>(N=xx) | EGT0001442<br>10 mg<br>(N=xx) | EGT0001442<br>20 mg<br>(N=xx) | EGT0001442<br>50 mg<br>(N=xx) |
| <br>Day 0 | Breakfast | n | XX | XX | XX | XX |
| | | Mean ± SD | xx.x ± x.xx | xx.x ± x.xx | xx.x ± x.xx | xx.x ± x.xx |
| | | Median | XX.X | XX.X | XX.X | XX.X |
| | | Min, Max | XX , XX | XX , XX | XX , XX | XX , XX |
| | Lunch | n | XX | XX | XX | XX |
| | 2411011 | Mean ± SD | xx.x ± x.xx | xx.x ± x.xx | xx.x ± x.xx | xx.x ± x.xx |
| | | Median | XX.X | XX.X | XX.X | XX.X |
| | | Min, Max | XX , XX | XX , XX | xx , xx | XX , XX |
| | Dinner | n | XX | XX | XX | XX |
| | DIMMEI | Mean ± SD | xx.x ± x.xx | xx.x ± x.xx | xx.x ± x.xx | xx.x ± x.xx |
| | | Median | XX.X | XX.X | XX.X | XX.X |
| | | Min, Max | XX , XX | XX , XX | XX , XX | XX , XX |
| ay 2 | Breakfast | n | XX XX | XX XX | XX | XX , XX |
| ay Z | DIEAKIASC | Mean ± SD | xx.x ± x.xx | xx.x ± x.xx | xx.x ± x.xx | xx.x ± x.xx |
| | | Median | XX.X | XX.X | XX.X | XX.X |
| | | Min, Max | | | | |
| | Lunch | • | xx , xx | xx , xx | xx , xx | xx , xx |
| | Lunch | n<br>Mean ± SD | XX 1 | XX | XX | XX 1 |
| | | | xx.x ± x.xx | xx.x ± x.xx | xx.x ± x.xx | xx.x ± x.xx |
| | | Median | XX.X | XX.X | XX.X | XX.X |
| | D. Lauren | Min, Max | XX , XX | xx , xx | XX , XX | xx , xx |
| | Dinner | n<br>Maran I OD | XX | XX | XX | XX |
| | | Mean ± SD | xx.x ± x.xx | xx.x ± x.xx | xx.x ± x.xx | xx.x ± x.xx |
| | | Median | XX.X | XX.X | XX.X | XX.X |
| | D 16 1 | Min, Max | xx , xx | XX , XX | XX , XX | XX , XX |
| hange from Day 0 | Breakfast | n<br>Maran I OD | XX | XX | XX | XX |
| o Day | | Mean ± SD | xx.x ± x.xx | xx.x ± x.xx | xx.x ± x.xx | xx.x ± x.xx |
| | | Median | XX.X | XX.X | XX.X | XX.X |
| | - 1 | Min, Max | xx , xx | XX , XX | XX , XX | XX , XX |
| | Lunch | n | XX | XX | XX | XX |
| | | Mean ± SD | $xx.x \pm x.xx$ | $xx.x \pm x.xx$ | xx.x ± x.xx | xx.x ± x.xx |
| | | Median | XX.X | XX.X | XX.X | XX.X |
| | | Min, Max | xx , xx | XX , XX | XX , XX | XX , XX |
| | Dinner | n | XX | XX | XX | XX |
| | | Mean ± SD | xx.x ± x.xx | $xx.x \pm x.xx$ | $xx.x \pm x.xx$ | xx.x ± x.xx |
| | | Median | XX.X | XX.X | XX.X | XX.X |
| | | Min, Max | xx , xx | xx , xx | xx , xx | xx , xx |

Table 14.2.16 Summary of Post Prandial Blood Glucose in AUC (mg.h/dL)

Dose Escalation Segment

| | | Dose Group | | | |
|---|---|---|---|---|---|
| | - | EGT0001442 | EGT0001442 | EGT0001442 | EGT0001442 |
| | | 5 mg | 10 mg | 20 mg | 50 mg |
| Day | Statistic | (N=XX) | (N=xx) | (N=xx) | (N=xx) |
| Day 0 | n | xx | xx | xx | xx |
| | Mean ± SD | xx.x ± x.xx | xx.x ± x.xx | xx.x ± x.xx | xx.x ± x.xx |
| | Median | xx.x | XX.X | XX.X | XX.X |
| | Min, Max | xx , xx | xx , xx | xx , xx | xx , xx |
| Day 2 | n | XX | XX | XX | XX |
| | Mean ± SD | $xx.x \pm x.xx$ | $xx.x \pm x.xx$ | $xx.x \pm x.xx$ | xx.x ± x.xx |
| | Median | XX.X | XX.X | XX.X | XX.X |
| | Min, Max | XX , XX | xx , xx | XX , XX | xx , xx |
| Change from Day 0 to Day 2 | n | XX | XX | XX | XX |
| | Mean ± SD | $xx.x \pm x.xx$ | $xx.x \pm x.xx$ | $xx.x \pm x.xx$ | $xx.x \pm x.xx$ |
| | Median | XX.X | XX.X | XX.X | XX.X |
| | Min, Max | xx , xx | xx , xx | xx , xx | xx , xx |

#### Table 14.3.1.1 Summary of TEAEs Double-blind Segment Double-blind Safety Analysis Set

Treatment Group

| | Placebo<br>(N=xx) | EGT0001442<br>5 mg<br>(N=xx) | EGT0001442<br>10 mg<br>(N=xx) | EGT0001442<br>20 mg<br>(N=xx) | EGT0001442<br>50 mg<br>(N=xx) |
|---|---|---|---|---|---|
| All TEAEs | xx ( xx.x%) E | xx ( xx.x%) E | xx ( xx.x%) E | xx ( xx.x%) E | xx ( xx.x%) E |
| Deaths | xx ( xx.x%) E | xx ( xx.x%) E | xx ( xx.x%) E | xx ( xx.x%) E | xx ( xx.x%) E |
| Serious TEAEs | xx ( xx.x%) E | xx ( xx.x%) E | xx ( xx.x%) E | xx ( xx.x%) E | xx ( xx.x%) E |
| TEAEs leading to withdrawal TEAEs related to study drug | xx ( xx.x%) E<br>xx ( xx.x%) E | xx ( xx.x%) E<br>xx ( xx.x%) E | xx ( xx.x%) E<br>xx ( xx.x%) E | xx ( xx.x%) E<br>xx ( xx.x%) E | xx ( xx.x%) E<br>xx ( xx.x%) E |

N: Number of subjects exposed in specified group

<sup>%:</sup> Percentage based on N

E: Number of TEAEs

## Table 14.3.1.2 Summary of TEAEs Dose Escalation Segment Dose Escalation Safety Analysis Set

| | Dose Group | | | |
|---|---|---|---|---|
| | EGT0001442 | EGT0001442 | EGT0001442 | EGT0001442 |
| | 5 mg | 10 mg | 20 mg | 50 mg |
| | (N=xx) | (N=xx) | (N=xx) | (N=xx) |
| All TEAEs Deaths Serious TEAEs TEAEs leading to study discontinuation TEAEs related to study drug | xx (xx.x%) E | xx (xx.x%) E | xx (xx.x%) E | xx ( xx.x%) E |
| | xx (xx.x%) E | xx (xx.x%) E | xx (xx.x%) E | xx ( xx.x%) E |

N: Number of subjects exposed in specified group

<sup>%:</sup> Percentage based on N

E: Number of TEAEs

Table 14.3.1.3 Summary of TEAEs by System Organ Class, Preferred Term and Treatment Group

Double-blind Segment

Double-blind Safety Analysis Set

| | Treatment Group | | | | |
|---|---|---|---|---|---|
| ystem Organ Class<br>Preferred Term | Placebo<br>(N=xx) | EGT0001442<br>5 mg<br>(N=xx) | EGT0001442<br>10 mg<br>(N=xx) | EGT0001442<br>20 mg<br>(N=xx) | EGT0001442<br>50 mg<br>(N=xx) |
| ubject with at least one AE | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| OC 1 | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| PT1 | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| PT2 | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| PTxx | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| OC 2 | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| PT1 | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx (xx.x%) |
| PT2 | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx (xx.x%) |
| PTxx | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |

Note: Counts reflect numbers of subjects reporting one or more adverse events that map to the MedDRA system organ class/preferred term. At each level of summarization (system organ class or preferred term), subjects reporting more than one adverse event are counted only once (under the greatest reported severity).

Note: N: Number of subjects in the specified group

%: Percentage based on N

#### Similar tables:

Table 14.3.1.4 Summary of Drug-related TEAEs by System Organ Class, Preferred Term and Treatment Group

Double-blind Segment

Double-blind Safety Analysis Set

Table 14.3.1.5 Summary of TEAEs Leading to Study Discontinuation by System Organ Class, Preferred Term and Treatment
Group
Double-blind Segment
Double-blind Safety Analysis Set

Table 14.3.1.6 Summary of Serious TEAEs by System Organ Class, Preferred Term and Treatment Group

Double-blind Segment

Double-blind Safety Analysis Set

Table 14.3.1.7 Summary of TEAEs by System Organ Class, Preferred Term and Dose Group

Dose Escalation Segment

Dose Escalation Safety Analysis Set

| | Dose Group | | | |
|---|---|---|---|---|
| System Organ Class<br>Preferred Term | EGT0001442<br>5 mg<br>(N=xx) | EGT0001442<br>10 mg<br>(N=xx) | EGT0001442<br>20 mg<br>(N=xx) | EGT0001442<br>50 mg<br>(N=xx) |
| ubject with at least one AE | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| OC 1 | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| PT1 | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| PT2 | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| PTxx | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| OC 2 | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| PT1 | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| PT2 | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| PTxx | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| OC 3 | | | | |

Note: Counts reflect numbers of subjects reporting one or more adverse events that map to the MedDRA system organ class/preferred term. At each level of summarization (system organ class or preferred term), subjects reporting more than one adverse event are counted only once (under the greatest reported severity).

Note: N: Number of subjects in the specified group

%: Percentage based on N

#### Similar tables:

Table 14.3.1.8 Summary of Drug-related TEAEs by System Organ Class, Preferred Term and Dose Group

Dose Escalation Segment

Dose Escalation Safety Analysis Set

Table 14.3.1.9 Summary of TEAEs Leading to Study Discontinuation by System Organ Class, Preferred Term and Dose Group

Dose Escalation Segment

Dose Escalation Safety Analysis Set

Table 14.3.1.10 Summary of Serious TEAEs by System Organ Class, Preferred Term and Dose Group

Dose Escalation Segment

Dose Escalation Safety Analysis Set

### Table 14.3.1.11 Summary of TEAEs by Maximum Severity Double-blind Segment Double-blind Safety Analysis Set

Treatment Group EGT0001442 EGT0001442 EGT0001442 EGT0001442 System Organ Class Placebo 5 mg 10 mg 20 mg 50 mg Preferred Term Severity (N=xx)(N=xx)(N=xx)(N=xx)(N=xx)Subject with at least one AE Mild xx (xx.x%) xx ( xx.x%) xx (xx.x%) xx (xx.x%) xx ( xx.x%) Moderate xx (xx.x%) xx (xx.x%)xx (xx.x%)xx (xx.x%)xx ( xx.x%) xx ( xx.x%) Severe xx (xx.x%) xx (xx.x%) xx (xx.x%) xx ( xx.x%) SOC 1 Mild xx (xx.x%) xx (xx.x%)xx ( xx.x%) xx (xx.x%)xx ( xx.x%) Moderate xx (xx.x%) xx (xx.x%) xx (xx.x%) xx ( xx.x%) xx (xx.x%) Severe xx (xx.x%) xx (xx.x%) xx (xx.x%) xx (xx.x%) xx (xx.x%) PT1 Mild xx (xx.x%) xx (xx.x%) xx (xx.x%) xx (xx.x%) xx (xx.x%) Moderate xx (xx.x%) xx (xx.x%) xx (xx.x%) xx (xx.x%) xx (xx.x%) Severe xx ( xx.x%) xx ( xx.x%) xx (xx.x%) xx (xx.x%) xx ( xx.x%) PTxx Mild xx (xx.x%) xx (xx.x%) xx (xx.x%) xx (xx.x%) xx ( xx.x%) Moderate xx (xx.x%)xx (xx.x%)xx (xx.x%)xx (xx.x%)xx ( xx.x%) Severe xx (xx.x%) xx (xx.x%) xx (xx.x%) xx (xx.x%) xx ( xx.x%) SOC 2 Mild xx (xx.x%)xx (xx.x%) xx (xx.x%)xx ( xx.x%) xx ( xx.x%) Moderate xx (xx.x%) xx (xx.x%) xx (xx.x%) xx (xx.x%) xx (xx.x%) Severe xx (xx.x%) xx (xx.x%) xx (xx.x%) xx (xx.x%) xx (xx.x%)

Note: Counts reflect numbers of subjects reporting one or more adverse events that map to the MedDRA system organ class/preferred term. At each level of summarization (system organ class or preferred term), subjects reporting more than one adverse event are counted only once (under the greatest reported severity).

Note: N: Number of subjects in the specified group

%: Percentage based on N

## Table 14.3.1.12 Summary of TEAEs by Maximum Severity Dose Escalation Segment Dose Escalation Safety Analysis Set

| | Treatment Group | | | | |
|---|---|---|---|---|---|
| System Organ Class<br>Preferred Term | Severity | EGT0001442<br>5 mg<br>(N=xx) | EGT0001442<br>10 mg<br>(N=xx) | EGT0001442<br>20 mg<br>(N=xx) | EGT0001442<br>50 mg<br>(N=xx) |
| Subject with at least one AE | Mild | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| | Moderate | xx (xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| | Severe | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| OC 1 | Mild | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| | Moderate | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| | Severe | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| PT1 | Mild | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| | Moderate | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| | Severe | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| PTxx | Mild | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| | Moderate | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| | Severe | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| SOC 2 | Mild | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| | Moderate | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| | Severe | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |

Note: Counts reflect numbers of subjects reporting one or more adverse events that map to the MedDRA system organ class/preferred term. At each level of summarization (system organ class or preferred term), subjects reporting more than one adverse event are counted only once (under the greatest reported severity).

Note: N: Number of subjects in the specified group

%: Percentage based on N

Table 14.3.1.13 Clinical Laboratory Evaluations in Biochemistry (Observed Values)

Double-blind Segment

Double-blind Safety Analysis Set

| | | | | | Treatment Group | | |
|---|---|---|---|---|---|---|---|
| | Visit<br>Day | Statistic | Placebo<br>(N=xx) | EGT0001442<br>5 mg<br>(N=xx) | EGT0001442<br>10 mg<br>(N=xx) | EGT0001442<br>20 mg<br>(N=xx) | EGT0001442<br>50 mg<br>(N=xx) |
| Albumin (G/L) | Screening | n | xx | XX | xx | xx | XX |
| (30 - 50) | 3 | Mean ± SD | xx.x ± x.xx | $xx.x \pm x.xx$ | $xx.x \pm x.xx$ | $xx.x \pm x.xx$ | xx.x ± x.xx |
| | | Median | xx.x | XX.X | XX.X | xx.x | XX.X |
| | | Min, Max | xx , xx | XX , XX | XX , XX | xx , xx | xx , xx |
| | Day -2 | n | XX | XX | XX | xx | XX |
| | | Mean ± SD | $xx.x \pm x.xx$ | $xx.x \pm x.xx$ | $xx.x \pm x.xx$ | $xx.x \pm x.xx$ | xx.x ± x.xx |
| | | Median | XX.X | XX.X | XX.X | XX.X | XX.X |
| | | Min, Max | xx , xx | XX , XX | XX , XX | xx , xx | XX , XX |
| | Day 1 | n | XX | XX | XX | XX | XX |
| | | Mean ± SD | $xx.x \pm x.xx$ | $xx.x \pm x.xx$ | $xx.x \pm x.xx$ | $xx.x \pm x.xx$ | xx.x ± x.xx |
| | | Median | XX.X | XX.X | XX.X | XX.X | XX.X |
| | | Min, Max | xx , xx | XX , XX | XX , XX | xx , xx | XX , XX |
| | • • • | | | | | | |
| ALT(SGPT) (U/L) | Screening | n | xx | xx | XX | xx | xx |
| (8 - 54) | | Mean ± SD | $xx.x \pm x.xx$ | $xx.x \pm x.xx$ | $xx.x \pm x.xx$ | $xx.x \pm x.xx$ | $xx.x \pm x.xx$ |
| | | Median | xx.x | XX.X | XX.X | XX.X | XX.X |
| | | Min, Max | XX , XX | xx , xx | xx , xx | xx , xx | xx , xx |

Note: Table will continue for other visit days 2, 8, 15, 22, 29, 35 and 43 and will continue for other lab parameters.

Table 14.3.1.14 Clinical Laboratory Evaluations in Change from Baseline in Biochemistry
Double-blind Segment
Double-blind Safety Analysis Set

| | | | | | Treatment Group | ) | |
|---|---|---|---|---|---|---|---|
| | Visit<br>Day | Statistic | Placebo<br>(N=xx) | EGT0001442<br>5 mg<br>(N=xx) | EGT0001442<br>10 mg<br>(N=xx) | EGT0001442<br>20 mg<br>(N=xx) | EGT0001442<br>50 mg<br>(N=xx) |
| Albumin (G/L)<br>(30 - 50) | Day 2 | n<br>Mean ± SD<br>Median<br>Min, Max<br>P-value* | xx<br>xx.x ± x.xx<br>xx.x<br>xx , xx<br>xx , xx | xx<br>xx.x ± x.xx<br>xx.x<br>xx , xx<br>xx , xx<br>x.xxxx | xx<br>xx.x ± x.xx<br>xx.x<br>xx , xx<br>xx , xx | xx<br>xx.x ± x.xx<br>xx.x<br>xx , xx<br>x.xxxx | xx<br>xx.x ± x.xx<br>xx.x<br>xx , xx<br>x.xxxx |
| | Day 8 | n<br>Mean ± SD<br>Median<br>Min, Max<br>P-value* | xx<br>xx.x ± x.xx<br>xx.x<br>xx , xx<br>x.xxxx | xx<br>xx.x ± x.xx<br>xx.x<br>xx , xx<br>x.xxxx | xx<br>xx.x ± x.xx<br>xx.x<br>xx , xx<br>xx , xx | xx<br>xx.x ± x.xx<br>xx.x<br>xx , xx<br>x.xxxx | xx<br>xx.x ± x.xx<br>xx.x<br>xx , xx<br>x.xxxx |
| ALT(SGPT) (U/L)<br>(8 - 54) | Day 2 | n<br>Mean ± SD<br>Median<br>Min, Max<br>P-value* | xx<br>xx.x ± x.xx<br>xx.x<br>xx , xx<br>x. , xx | xx<br>xx.x ± x.xx<br>xx.x<br>xx , xx<br>xx , xx | xx<br>xx.x ± x.xx<br>xx.x<br>xx , xx<br>xx , xx | xx<br>xx.x ± x.xx<br>xx.x<br>xx , xx<br>x.xxxx | xx<br>xx.x ± x.xx<br>xx.x<br>xx , xx<br>x.xxxx |

Note: Baseline is defined as the last observed measurement prior to dosing on Day 1 at Visit 5.

Note: \*P-values are from paired t-test.

Note: Table will continue for other visit days 15, 22, 29, 35 and 43 and will continue for other lab parameters.

Table 14.3.1.15 Biochemistry Laboratory Shift Table
Double-blind Segment
Double-blind Safety Analysis Set

| Lab<br>Parameter | | | | Day 1 / Baseline | | | | |
|---|---|---|---|---|---|---|---|---|
| | Treatment | Visit<br>Day | _ | Missing<br>n (%) | Below LLNR n (%) | Normal<br>n (%) | Above ULNR<br>n (%) | Total<br>n (%) |
| Albumin (G/L) (30 - 50) | Placebo (N=xx) | Day 2 | Missing<br>Below LLNR<br>Normal<br>Above ULNR<br>Total | xx ( xx.x)<br>xx ( xx.x)<br>xx ( xx.x)<br>xx ( xx.x)<br>xx ( xx.x) | xx ( xx.x)<br>xx ( xx.x)<br>xx ( xx.x)<br>xx ( xx.x)<br>xx ( xx.x) | xx ( xx.x)<br>xx ( xx.x)<br>xx ( xx.x)<br>xx ( xx.x)<br>xx ( xx.x) | xx ( xx.x)<br>xx ( xx.x)<br>xx ( xx.x)<br>xx ( xx.x)<br>xx ( xx.x) | xx ( xx.x)<br>xx ( xx.x)<br>xx ( xx.x)<br>xx ( xx.x)<br>xx ( xx.x)<br>xx (100.0) |
| | | Day 8 | Missing<br>Below LLNR<br>Normal<br>Above ULNR<br>Total | xx ( xx.x)<br>xx ( xx.x)<br>xx ( xx.x)<br>xx ( xx.x)<br>xx ( xx.x) | xx ( xx.x)<br>xx ( xx.x)<br>xx ( xx.x)<br>xx ( xx.x)<br>xx ( xx.x) | xx ( xx.x)<br>xx ( xx.x)<br>xx ( xx.x)<br>xx ( xx.x)<br>xx ( xx.x) | xx ( xx.x)<br>xx ( xx.x)<br>xx ( xx.x)<br>xx ( xx.x)<br>xx ( xx.x) | xx (xx.x)<br>xx (xx.x)<br>xx (xx.x)<br>xx (xx.x)<br>xx (100.0) |

EGT0001442 5 mg (N=xx)

. . .

Note: N: Number of subjects in the specified group

n: Number subjects with data available

%: Percentage based on N

LLNR: Lower Limit of Normal Range ULNR: Upper Limit of Normal Range

Table will continue for other visit days 15, 22, 29, 35 and 43 and for other treatment group and other lab parameters.

#### Similar tables:

Table 14.3.1.16 Clinical Laboratory Evaluations in Hematology (Observed Values)

Double-blind Segment

Double-blind Safety Analysis Set

Table 14.3.1.17 Clinical Laboratory Evaluations in Change from Baseline in Hematology
Double-blind Segment
Double-blind Safety Analysis Set

Table 14.3.1.18 Hematology Laboratory Shift Table
Double-blind Segment
Double-blind Safety Analysis Set

Table 14.3.1.19 Clinical Laboratory Evaluations in Urinalysis (Observed Values)

Double-blind Segment

Double-blind Safety Analysis Set

Table 14.3.1.20 Clinical Laboratory Evaluations in Change from Baseline in Urinalysis

Double-blind Segment

Double-blind Safety Analysis Set

## Table 14.3.1.21 Urinalysis Laboratory Shift Table Double-blind Segment Double-blind Safety Analysis Set

| | | | | | Day 1 / | Baseline | |
|---|---|---|---|---|---|---|---|
| Lab<br>Parameter | Treatment | Visit<br>Day | - | Missing<br>n (%) | Normal<br>n (%) | Abnormal n (%) | Total<br>n (%) |
| lbumin (G/L) | Placebo (N=xx) | Day 2 | Missing | xx ( xx.x) | xx ( xx.x) | xx ( xx.x) | xx ( xx.x) |
| 30 - 50) | | | Normal<br>Abnormal | xx ( xx.x) | xx ( xx.x) | xx ( xx.x) | xx ( xx.x) |
| | | | Total | xx ( xx.x)<br>xx ( xx.x) | xx ( xx.x)<br>xx ( xx.x) | xx ( xx.x)<br>xx ( xx.x) | xx ( xx.x)<br>xx (100.0) |
| | | Day 8 | Missing | xx ( xx.x) | xx ( xx.x) | xx ( xx.x) | xx ( xx.x) |
| | | - 2 | Normal | xx (xx.x) | xx ( xx.x) | xx ( xx.x) | xx ( xx.x) |
| | | | Abnormal | xx ( xx.x) | xx ( xx.x) | xx ( xx.x) | xx ( xx.x) |
| | | | Total | xx ( xx.x) | xx ( xx.x) | xx ( xx.x) | xx (100.0) |

Note: N: Number of subjects in the specified group

n: Number subjects with data available

%: Percentage based on N

Table will continue for other visit days 15, 22, 29, 35 and 43 and for other treatment group and other lab parameters.

Table 14.3.1.22 Clinical Laboratory Evaluations in Biochemistry (Observed Values)

Dose Escalation Segment

Dose Escalation Safety Analysis Set

| | Visit | | Dose Group | | | |
|---|---|---|---|---|---|---|
| | | | EGT0001442<br>5 mg | | EGT0001442 | EGT0001442 |
| | Day | Statistic | (N=xx) | (N=xx) | (N=xx) | (N=xx) |
| lbumin (G/L) | Screening | n | xx | XX | xx | xx |
| 30 - 50) | | Mean ± SD | xx.x ± x.xx | xx.x ± x.xx | xx.x ± x.xx | xx.x ± x.xx |
| • | | Median | xx.x | XX.X | XX.X | XX.X |
| | | Min, Max | xx , xx | xx , xx | XX , XX | xx , xx |
| | Day 0 | n | xx | XX | XX | XX |
| | | Mean ± SD | $xx.x \pm x.xx$ | $xx.x \pm x.xx$ | $xx.x \pm x.xx$ | $xx.x \pm x.xx$ |
| | | Median | XX.X | XX.X | XX.X | XX.X |
| | | Min, Max | xx , xx | xx , xx | XX , XX | XX , XX |
| | Day 1 | n | XX | XX | XX | XX |
| | | Mean ± SD | $xx.x \pm x.xx$ | $xx.x \pm x.xx$ | $xx.x \pm x.xx$ | $xx.x \pm x.xx$ |
| | | Median | XX.X | XX.X | XX.X | XX.X |
| | | Min, Max | XX , XX | xx , xx | XX , XX | XX , XX |
| | • • • | | | | | |
| LT(SGPT) (U/L) | Screening | n | xx | xx | xx | xx |
| 3 - 54) | | Mean ± SD | $xx.x \pm x.xx$ | $xx.x \pm x.xx$ | xx.x ± x.xx | $xx.x \pm x.xx$ |
| | | Median | xx.x | XX.X | XX.X | XX.X |
| | | Min, Max | xx , xx | xx , xx | xx , xx | XX , XX |

Note: Table will continue for other visit days 2, 3, 8, 15, 22, 23 and 43 and will continue for other lab parameters.

Similar tables:

Table 14.3.1.23 Clinical Laboratory Evaluations in Hematology (Observed Values)

Dose Escalation Segment

Dose Escalation Safety Analysis Set

Table 14.3.1.24 Clinical Laboratory Evaluations in Urinalysis (Observed Values)

Dose Escalation Segment

Dose Escalation Safety Analysis Set

Table 14.3.1.25 Summary of Vital Signs (Observed Values)
Double-blind Segment
Double-blind Safety Analysis Set

| | | | | | Treatment Group | | |
|---|---|---|---|---|---|---|---|
| | Visit<br>Day | Statistic | Placebo<br>(N=xx) | EGT0001442<br>5 mg<br>(N=xx) | EGT0001442<br>10 mg<br>(N=xx) | EGT0001442<br>20 mg<br>(N=xx) | EGT0001442<br>50 mg<br>(N=xx) |
| Pulse (beats/minute) | Screening | n<br>Mean ± SD<br>Median<br>Min, Max | xx<br>xx.x ± x.xx<br>xx.x<br>xx , xx | xx<br>xx.x ± x.xx<br>xx.x<br>xx , xx | xx<br>xx.x ± x.xx<br>xx.x<br>xx , xx | xx<br>xx.x ± x.xx<br>xx.x<br>xx , xx | xx<br>xx.x ± x.xx<br>xx.x<br>xx , xx |
| | Day -2 | n<br>Mean ± SD<br>Median<br>Min, Max | xx , xx ± x.xx xx .x , xx | xx '<br>xx.x ± x.xx<br>xx.x<br>xx , xx | xx , xx ± x.xx xx.x xx , xx | xx<br>xx.x ± x.xx<br>xx.x<br>xx , xx | xx , xx ± x.xx xx.x xx , xx |
| | Day 1/Pre-dose | n<br>Mean ± SD<br>Median<br>Min, Max | xx<br>xx.x ± x.xx<br>xx.x<br>xx.x | xx<br>xx.x ± x.xx<br>xx.x<br>xx , xx | xx<br>xx.x ± x.xx<br>xx.x<br>xx , xx | xx<br>xx.x ± x.xx<br>xx.x<br>xx , xx | xx<br>xx.x ± x.xx<br>xx.x<br>xx , xx |
| | Day 2/Pre-dose Day 8 Day 15 Day 22 Day 29 Day 35 Day 43 | , | · | , | , | • | · |
| Systolic BP (mmHg) | Screening | n<br>Mean ± SD<br>Median<br>Min, Max | xx<br>xx.x ± x.xx<br>xx.x<br>xx , xx | xx<br>xx.x ± x.xx<br>xx.x<br>xx , xx | xx<br>xx.x ± x.xx<br>xx.x<br>xx , xx | xx<br>xx.x ± x.xx<br>xx.x<br>xx , xx | xx<br>xx.x ± x.xx<br>xx.x<br>xx , xx |

Note: Table will continue for other vital signs.

Table 14.3.1.26 Summary of Vital Signs in Change from Baseline Double-blind Segment Double-blind Safety Analysis Set

| | | | | | Treatment Group | | |
|---|---|---|---|---|---|---|---|
| | Visit<br>Day | Statistic | Placebo<br>(N=xx) | EGT0001442<br>5 mg<br>(N=xx) | EGT0001442<br>10 mg<br>(N=xx) | EGT0001442<br>20 mg<br>(N=xx) | EGT0001442<br>50 mg<br>(N=xx) |
| Pulse (beats/minute) | Day 2 | n<br>Mean ± SD<br>Median<br>Min, Max<br>P-value* | xx<br>xx.x ± x.xx<br>xx.x<br>xx , xx<br>xx , xx | xx<br>xx.x ± x.xx<br>xx.x<br>xx , xx<br>xx , xx<br>x.xxxx | xx<br>xx.x ± x.xx<br>xx.x<br>xx , xx<br>xx , xx | xx<br>xx.x ± x.xx<br>xx.x<br>xx , xx<br>x.xxxx | xx<br>xx.x ± x.xx<br>xx.x<br>xx , xx<br>x.xxxx |
| | Day 8 | n<br>Mean ± SD<br>Median<br>Min, Max<br>P-value* | xx<br>xx.x ± x.xx<br>xx.x<br>xx , xx<br>x.xxxx | xx<br>xx.x ± x.xx<br>xx.x<br>xx , xx<br>x.xxxx | xx<br>xx.x ± x.xx<br>xx.x<br>xx , xx<br>x.xxxx | xx<br>xx.x ± x.xx<br>xx.x<br>xx , xx<br>x.xxxx | xx<br>xx.x ± x.xx<br>xx.x<br>xx , xx<br>x.xxxx |
| ystolic BP (mmHq) | Day 2 | n | XX | xx | xx | xx | xx |
| ,000110 <i>D1</i> (mming) | 24, 2 | Mean ± SD<br>Median<br>Min, Max<br>P-value* | xx.x ± x.xx<br>xx.x<br>xx , xx<br>xx , xx | xx.x ± x.xx<br>xx.x<br>xx , xx<br>xx , xx | xx.x ± x.xx<br>xx.x<br>xx , xx<br>xx , xx | xx.x ± x.xx<br>xx.x<br>xx , xx<br>xx , xx<br>x.xxxx | xx.x ± x.xx<br>xx.x<br>xx , xx<br>xx , xx |

Note: Baseline is defined as the last observed measurement prior to dosing on Day 1 at Visit 5.

Note: \*P-values are from paired t-test.

Note: Table will continue for other days 8, 15, 22, 29, 35 and 43 and will continue for other vital signs.

Table 14.3.1.27 Summary of Vital Signs (Observed Values)
Dose Escalation Segment
Dose Escalation Safety Analysis Set

| | | | Dose Group | | | |
|---|---|---|---|---|---|---|
| | Visit<br>Day Stati | stic | EGT0001442<br>5 mg<br>(N=xx) | EGT0001442<br>10 mg<br>(N=xx) | EGT0001442<br>20 mg<br>(N=xx) | EGT0001442<br>50 mg<br>(N=xx) |
| ulse (beats/minute) | Screening | n<br>Mean ± SD<br>Median<br>Min, Max | xx<br>xx.x ± x.xx<br>xx.x<br>xx.x | xx<br>xx.x ± x.xx<br>xx.x<br>xx , xx | xx<br>xx.x ± x.xx<br>xx.x<br>xx , xx | xx<br>xx.x ± x.xx<br>xx.x<br>xx , xx |
| | Day 0 | n<br>Mean ± SD<br>Median<br>Min, Max | xx.x ± x.xx<br>xx.x<br>xx.x<br>xx.x | xx xx ± x.xx xx.x xx.x xx.x | xx xx ± x.xx xx.x xx.x xx.x | xx<br>xx.x ± x.xx<br>xx.x<br>xx , xx |
| | Day 1/Pre-dose | n<br>Mean ± SD<br>Median<br>Min, Max | xx<br>xx.x ± x.xx<br>xx.x<br>xx , xx | xx<br>xx.x ± x.xx<br>xx.x<br>xx , xx | xx<br>xx.x ± x.xx<br>xx.x<br>xx , xx | xx<br>xx.x ± x.xx<br>xx.x<br>xx , xx |
| | Day 1/1 hr Day 1/2 hr Day 1/4 hr Day 1/8 hr Day 2/Pre-dose Day 3/Pre-dose Day 8 Day 15 Day 22 Day 29 Day 43 | | | | | |

Note: Table will continue for other vital signs

# Table 14.3.1.28 Summary of 12-Lead ECG (Observed Values) Double-blind Segment Double-blind Safety Analysis Set

| | | | | | Treatment Group | | |
|---|---|---|---|---|---|---|---|
| | Visit<br>Day | Statistic | Placebo<br>(N=xx) | EGT0001442<br>5 mg<br>(N=xx) | EGT0001442<br>10 mg<br>(N=xx) | EGT0001442<br>20 mg<br>(N=xx) | EGT0001442<br>50 mg<br>(N=xx) |
| PR Interval (ms) | Screening | n<br>Mean ± SD<br>Median<br>Min, Max | xx<br>xx.x ± x.xx<br>xx.x<br>xx , xx | xx<br>xx.x ± x.xx<br>xx.x<br>xx , xx | xx<br>xx.x ± x.xx<br>xx.x<br>xx , xx | xx<br>xx.x ± x.xx<br>xx.x<br>xx , xx | xx<br>xx.x ± x.xx<br>xx.x<br>xx , xx |
| | Day -2 | n<br>Mean ± SD<br>Median<br>Min, Max | xx<br>xx.x ± x.xx<br>xx.x<br>xx.x | xx<br>xx.x ± x.xx<br>xx.x<br>xx.x | xx xx.x ± x.xx xx.x xx.x | xx<br>xx.x ± x.xx<br>xx.x<br>xx.x | xx<br>xx.x ± x.xx<br>xx.x<br>xx.x |
| | Day 1/Pre-dose | n<br>Mean ± SD<br>Median<br>Min, Max | xx<br>xx.x ± x.xx<br>xx.x<br>xx.x | xx<br>xx.x ± x.xx<br>xx.x<br>xx , xx | xx<br>xx.x ± x.xx<br>xx.x<br>xx , xx | xx<br>xx.x ± x.xx<br>xx.x<br>xx.x | xx<br>xx.x ± x.xx<br>xx.x<br>xx , xx |
| | Day 29 | | | | | | |
| QRS Interval (ms) | Screening | n<br>Mean ± SD<br>Median<br>Min, Max | xx<br>xx.x ± x.xx<br>xx.x<br>xx , xx | xx<br>xx.x ± x.xx<br>xx.x<br>xx , xx | xx<br>xx.x ± x.xx<br>xx.x<br>xx , xx | xx<br>xx.x ± x.xx<br>xx.x<br>xx , xx | xx<br>xx.x ± x.xx<br>xx.x<br>xx , xx |

Note: Table will continue for other ECGs.

Table 14.3.1.29 Summary of 12-Lead ECG in Change from Baseline
Double-blind Segment
Double-blind Safety Analysis Set

| | | | | Treatment Group | | |
|---|---|---|---|---|---|---|
| Visit<br>Day | Statistic | Placebo<br>(N=xx) | EGT0001442<br>5 mg<br>(N=xx) | EGT0001442<br>10 mg<br>(N=xx) | EGT0001442<br>20 mg<br>(N=xx) | EGT0001442<br>50 mg<br>(N=xx) |
| Day 2 | n<br>Mean ± SD<br>Median<br>Min, Max<br>P-value* | xx<br>xx.x ± x.xx<br>xx.x<br>xx , xx<br>xx , xx | xx<br>xx.x ± x.xx<br>xx.x<br>xx , xx<br>xx , xx<br>x.xxxx | xx<br>xx.x ± x.xx<br>xx.x<br>xx , xx<br>xx , xx<br>x.xxxx | xx<br>xx.x ± x.xx<br>xx.x<br>xx , xx<br>x.xxxx | xx<br>xx.x ± x.xx<br>xx.x<br>xx , xx<br>x.xxxx |
| Day 8 | n<br>Mean ± SD<br>Median<br>Min, Max<br>P-value* | xx<br>xx.x ± x.xx<br>xx.x<br>xx , xx<br>x.xxxx | xx<br>xx.x ± x.xx<br>xx.x<br>xx , xx<br>x.xxxx | xx<br>xx.x ± x.xx<br>xx.x<br>xx , xx<br>x.xxxx | xx<br>xx.x ± x.xx<br>xx.x<br>xx , xx<br>x.xxxx | xx<br>xx.x ± x.xx<br>xx.x<br>xx , xx<br>x.xxxx |
| Day 2 | n<br>Mean ± SD<br>Median<br>Min, Max<br>P-value* | xx<br>xx.x ± x.xx<br>xx.x<br>xx , xx<br>x.xxxx | xx<br>xx.x ± x.xx<br>xx.x<br>xx , xx<br>x.xxxx | xx<br>xx.x ± x.xx<br>xx.x<br>xx , xx<br>x.xxxx | xx<br>xx.x ± x.xx<br>xx.x<br>xx , xx<br>x.xxxx | xx<br>xx.x ± x.xx<br>xx.x<br>xx , xx<br>x.xxxx |
| | Day 2 Day 8 | Day 2 n Mean ± SD Median Min, Max P-value* Day 8 n Mean ± SD Median Min, Max P-value* Day 2 n Mean ± SD Median Min, Max P-value* | Day 2 | Visit Placebo 5 mg (N=xx) Day 2 n xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx <td>Visit Day Day Statistic Day 2 Day 2 Day 2 Day 3 Day 3 Day 4 Day 5 Day 6 Day 6 Day 6 Day 6 Day 6 Day 7 Day 7 Day 8 Day 8 Day 8 Day 8 Day 8 Day 8 Day 8 Day 8 Day 8 Day 9 Day 9 Day 9 Day 9 Day 9 Day 9 Day 9 Day 9 Day 9 Day 9 Day 9 Day 9 Day 9 Day 9 Day 9 Day 9 Day 9 Day 9 Day 9 Day 9 Day 9 Day 9 Day 9 Day 9 Day 9 Day 9 Day 9 Day 9 Day 9 Day 9 Day 9 Day 9 Day 9 Day 9 Day 9 Day 9 Day 9 Day 9 Day 9 Day 9 Day 9 Day 1 Day 1 Day 1 Day 1 Day 1 Day 1 Day 1 Day 2 Day 1 Day 2 Day 1 Day 2 Day 1 Day 1 Day 1 Day 2 Day 1 Day 2 Day 1 Day 2 Day 1 Day 2 Day 1 Day 2 Day 2 Day 1 Day 2 Day 2 Day 1 Day 2 Day 2 Day 2 Day 1 Day 2 Day 2 Day 2 Day 2 Day 2 Day 2 Day 2 Day 3 Day 2 Day 2 Day 2 Day 2 Day 3 Day 3 Day 3 Day 3 Day 4 Day 4 Day 4 Day 4 Day 7 Day 8 Day 7 Day 8 Day 8 Day 8 Day 8 Day 8 Day 9 Day 8 Day 8 Day 9 Day 9 Day 1 Day 8 Day 1 Day 8 Day 1 Day 8 Day 1 Day 8 Day 1 Day 8 Day 1 Day 8 Day 1 Day 8 Day 1 Day 8 Day 1 Day 8 Day 1 Day 8 Day 1 Day 1 Day 8 Day 1 Day 1 Day 1 Day 1 Day 1 Day 1 Day 1 Day 1 Day 1 Day 1 Day 1 Day 1 Day 1 Day 1 Day 1 Day 1 Day 1 Day 1 Day 1 Day 1 Day 1 Day 1 Day 1 Day 1 Day 1 Day 1 Day 1 Day 1 Day 1 Day 1 Day 1 Day 1 Day 1 Day 1 Day 1 Day 1 Day 1 Day 1 Day 1 Day 1 Day 1 Day 1 Day 1 Day 1 Day 1 Day 1 Day 1 Day 1 Day 1 Day 1 Day 1 Day 1 Day 1 Day 1 Day 1 Day 1 Day 1 Day 1 Day 1 Day 1 Day 1 Day 1 Day 1 Day 1 Day 1 Day 1 Day 1 Day 1 Day 1 Day 1 Day 1 Day 1 Day 1 Day 1 Day 1 Day 1 Day 1 Day 1 Day 1 Day 1 Day 1 Day 1 Day 1 Day 1 Day 1 Day 1 Day 1 Day 1 Day 1 Day 1 Day 1 Day 1 Day 1 Day 1 Day 1 Day 1 Day 1 Day 1 Day 1 Day 1 Day 1 Day 1 Day 1 Day 1 Day 1 Day 1 Day 1 Day 1 Day 1 Day 1 Day 1 Day 1 Day 1 Day 1 Day 1 Day 1 Day 1 Day 1 Day 1 Day 1 Day 1 Day 1 Day 1 Day 1 Day 1 Day 1 Day 1 Day 1 Day 1 Day 1 Day 1 Day 1 Day 1 Day 1 Day</td> <td>Visit Day Statistic Placebo (N=xx) 5 mg (N=xx) 10 mg (N=xx) 20 mg (N=xx) Day 2 n xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx</td> | Visit Day Day Statistic Day 2 Day 2 Day 2 Day 3 Day 3 Day 4 Day 5 Day 6 Day 6 Day 6 Day 6 Day 6 Day 7 Day 7 Day 8 Day 9 Day 1 Day 1 Day 1 Day 1 Day 1 Day 1 Day 1 Day 2 Day 1 Day 2 Day 1 Day 2 Day 1 Day 1 Day 1 Day 2 Day 1 Day 2 Day 1 Day 2 Day 1 Day 2 Day 1 Day 2 Day 2 Day 1 Day 2 Day 2 Day 1 Day 2 Day 2 Day 2 Day 1 Day 2 Day 2 Day 2 Day 2 Day 2 Day 2 Day 2 Day 3 Day 2 Day 2 Day 2 Day 2 Day 3 Day 3 Day 3 Day 3 Day 4 Day 4 Day 4 Day 4 Day 7 Day 8 Day 7 Day 8 Day 8 Day 8 Day 8 Day 8 Day 9 Day 8 Day 8 Day 9 Day 9 Day 1 Day 8 Day 1 Day 1 Day 8 Day 1 Day | Visit Day Statistic Placebo (N=xx) 5 mg (N=xx) 10 mg (N=xx) 20 mg (N=xx) Day 2 n xx xx |

Note: Baseline is defined as the last observed measurement prior to dosing on Day 1 at Visit 5.

Note: \*P-values are from paired t-test.

Note: Table will continue for other days 15, 22 and 29 and will continue for other ECGs.

## Table 14.3.1.30 Summary of 12-Lead ECG (Observed Values) Dose Escalation Segment Dose Escalation Safety Analysis Set

Dose Group EGT0001442 EGT0001442 EGT0001442 EGT0001442 Visit 5 mg 10 mg 20 mg 50 mg Day Statistic (N=xx)(N=xx)(N=xx)(N=xx)Pulse (beats/minute) Screening Mean ± SD  $xx.x \pm x.xx$ xx.x ± x.xx  $xx.x \pm x.xx$  $xx.x \pm x.xx$ Median XX.X XX.X XX.X XX.X Min, Max XX , XX XX , XX XX , XX xx , xx Day 0 XX Mean ± SD  $xx.x \pm x.xx$  $xx.x \pm x.xx$  $xx.x \pm x.xx$ xx.x ± x.xx Median XX.X XX.X XX.X XX.X Min, Max xx , xx xx , xx xx , xx xx , xx Day 1/Pre-dose XX XX XX XX Mean ± SD  $xx.x \pm x.xx$  $xx.x \pm x.xx$  $xx.x \pm x.xx$  $xx.x \pm x.xx$ Median XX.X XX.X XX.X XX.X Min, Max XX , XX XX , XX xx , xx XX , XX Day 1/2 hr Day 2/Pre-dose Day 29 Systolic BP (mmHg) Screening Mean ± SD  $xx.x \pm x.xx$  $xx.x \pm x.xx$  $xx.x \pm x.xx$  $xx.x \pm x.xx$ Median XX.X XX.X XX.X XX.X Min, Max xx , xx xx , xx xx , xx xx , xx

Note: Table will continue for other ECGs.

Table 14.3.1.31 Summary of Fasting Plasma Glucose by Visit (Observed Values)

Double-blind Segment

Double-blind Safety Analysis Set

| | | Treatment Group | | | | |
|---|---|---|---|---|---|---|
| Visit<br>Day | Statistic | Placebo<br>(N=xx) | EGT0001442<br>5 mg<br>(N=xx) | EGT0001442<br>10 mg<br>(N=xx) | EGT0001442<br>20 mg<br>(N=xx) | EGT0001442<br>50 mg<br>(N=xx) |
| Screening | n | XX | XX | xx | XX | XX |
| | Mean ± SD | xx.x ± x.xx | xx.x ± x.xx | $xx.x \pm x.xx$ | $xx.x \pm x.xx$ | xx.x ± x.xx |
| | Median | xx.x | XX.X | xx.x | XX.X | XX.X |
| | Min, Max | XX , XX | xx , xx | XX , XX | XX , XX | xx , xx |
| ay -2 | n | XX | xx | XX | XX | xx |
| _ | Mean ± SD | xx.x ± x.xx | xx.x ± x.xx | $xx.x \pm x.xx$ | $xx.x \pm x.xx$ | xx.x ± x.xx |
| | Median | xx.x | XX.X | xx.x | XX.X | XX.X |
| | Min, Max | XX , XX | xx , xx | XX , XX | XX , XX | xx , xx |
| ay 1 | n | XX | xx | XX | XX | xx |
| | Mean ± SD | xx.x ± x.xx | $xx.x \pm x.xx$ | $xx.x \pm x.xx$ | $xx.x \pm x.xx$ | $xx.x \pm x.xx$ |
| | Median | XX.X | XX.X | XX.X | XX.X | XX.X |
| | Min, Max | XX , XX | xx , xx | XX , XX | XX , XX | xx , xx |

Note: Table will continue for Days 2,8,15,22,27,29,35,41 and 43.

### Table 14.3.1.32 Summary of Concomitant Medication Double-blind Segment Double-blind Safety Analysis Set

Treatment Group EGT0001442 EGT0001442 EGT0001442 EGT0001442 Placebo 5 mg 10 mg 20 mg 50 mg Preferred Medication Term (N=xx)(N=xx)(N=xx)(N=xx)(N=xx)Any Medication xx (xx.x%) xx (xx.x%) xx ( xx.x%) xx ( xx.x%) xx (xx.x%) ConMed 1 xx (xx.x%) xx ( xx.x%) xx ( xx.x%) xx ( xx.x%) xx (xx.x%) ConMed 2 xx ( xx.x%) xx ( xx.x%) xx ( xx.x%) xx ( xx.x%) xx (xx.x%) ConMed 3 xx (xx.x%) xx ( xx.x%) xx ( xx.x%) xx ( xx.x%) xx (xx.x%) ConMed 4 xx ( xx.x%) xx ( xx.x%) xx ( xx.x%) xx ( xx.x%) xx (xx.x%)

Note: A subject is counted only once per concomitant medication.

N: Number of subjects exposed

<sup>%:</sup> Percentage is based N

## Table 14.3.1.33 Summary of Concomitant Medication Dose Escalation Segment Dose Escalation Safety Analysis Set

Dose Group EGT0001442 EGT0001442 EGT0001442 EGT0001442 5 mg 10 mg 20 mg 50 mg Preferred Medication Term (N=xx)(N=xx)(N=xx)(N=xx)Any Medication xx (xx.x%) xx ( xx.x%) xx ( xx.x%) xx ( xx.x%) ConMed 1 xx ( xx.x%) xx ( xx.x%) xx (xx.x%) xx ( xx.x%) ConMed 2 xx ( xx.x%) xx ( xx.x%) xx ( xx.x%) xx ( xx.x%) ConMed 3 xx ( xx.x%) xx ( xx.x%) xx ( xx.x%) xx ( xx.x%) ConMed 4 xx ( xx.x%) xx ( xx.x%) xx ( xx.x%) xx (xx.x%)

Note: A subject is counted only once per concomitant medication.

N: Number of subjects in the specified group

%: Percentage is based N

#### **Summary Listings**

Listing 16.2.1 Subject Disposition

| Study<br>Segment | Treatment | Center | Subject<br>Number | Date<br>Last/<br>Contact | Termination<br>Status | Termination<br>Reason |
|---|---|---|---|---|---|---|
| Double-blind | Placebo | 02 | 02141<br>02142 | ddmmmyyyy<br>ddmmmyyyy | Completed<br>Discontinued due to adverse event | ******* |
| | | ••• | | | | |
| | EGT0001442 5 mg | | | | | |
| | EGT0001442 10 mg | | | | | |
| | EGT0001442 20 mg | | | | | |
| | EGT0001442 50 mg | | | | | |
| Dose Escalation | EGT0001442 5 mg | 01 | 003 | ddmmmyyyy | Completed | |
| | EGT0001442 10 mg | ••• | | | | |
| | EGT0001442 20 mg | | | | | |
| | EGT0001442 50 mg | | | | | |

#### Listing 16.2.2 Protocol Deviations

| Study<br>Segment | Treatment | Center | Subject<br>Number | Deviation<br>Date /Time | Page ID | Deviation<br>Category | Description of<br>Deviation | Deviation<br>Major/minor |
|---|---|---|---|---|---|---|---|---|
| Double-blind | Placebo | 02 | 02141 | ddmmmyyyy/hhmm | EX0012 | DOSING | xxxxxxxxxxx | Minor |
| | | • • • | | | | | | |
| | EGT0001442 5 | mg | | | | | | |
| | EGT0001442 10 | ) mg | | | | | | |
| | EGT0001442 20 | ) mg | | | | | | |
| | EGT0001442 50 | ) mg | | | | | | |
| Dose Escalation | EGT0001442 5 | mg 0 | 1 003 | ddmmmyyyy/hhmm | EX0012 | DOSING | xxxxxxxxxxx | NA |
| | EGT0001442 10 | ) mg | | | | | | |
| | EGT0001442 20 | ) mg | | | | | | |
| | EGT0001442 50 | ) ma | | | | | | |

#### Listing 16.2.3 Subjects Excluded from the Efficacy Analysis (Double-blind Segment)

| Treatment | Center | Subject<br>Number | Safety Population | ITT Population | PP Population |
|---|---|---|---|---|---|
| Placebo | 02 | 02141 | Yes | No | No |

EGT0001442 5 mg

EGT0001442 10 mg

EGT0001442 20 mg

EGT0001442 50 mg

#### Listing 16.2.4.1 Demographics

| Study<br>Segment | Treatment | Center | Subject<br>Number | Date of<br>Birth | Age<br>(yrs) | Gender | Race | Ethnicity | Height<br>(cm) | Weight<br>(kg) | BMI<br>(kg/m^2) |
|---|---|---|---|---|---|---|---|---|---|---|---|
| Double-blind | Placebo | 02 | 02141 | ddmmmyyyy | XX | Male | White | Hispanic or Latino | XXX | xxx.x | xxx.x |
| | EGT0001442 | 5 mg | | | | | | | | | |
| | EGT0001442 | 10 mg | | | | | | | | | |
| | EGT0001442 | 20 mg | | | | | | | | | |
| | EGT0001442 | 50 mg | | | | | | | | | |
| Dose Escalation | EGT0001442 | 5 mg | | | | | | | | | |
| | EGT0001442 | 10 mg | | | | | | | | | |
| | EGT0001442 | 20 mg | | | | | | | | | |
| | EGT0001442 | 50 mg | | | | | | | | | |
# Listing 16.2.4.2 Medical History

| Study<br>Segment | Treatment | Center | Subject<br>Number | Seq.<br>No. | Body<br>System | Medical history<br>Findings | Start<br>Date | Ongoing | Stop<br>Date |
|---|---|---|---|---|---|---|---|---|---|
| Double-blind | Placebo | 02 | 02141 | 1<br>2<br>3<br>4 | Eyes, Ears, Nose, Throat<br>Neurological<br>Cardiovascular<br>Skin | NORMAL<br>OCCASIONAL HEADACHES<br>HIGH CHOLESTEROL<br>BALANITIS | UNKUNK1989<br>UNKUNK2007<br>21DEC2009 | Yes<br>Yes | 29DEC2009 |
| | | | | • • • | | | | | |
| | | • • • | | | | | | | |
| | EGT0001442 | 5 mg | | | | | | | |
| | EGT0001442 | 10 mg | | | | | | | |
| | EGT0001442 | 20 mg | | | | | | | |
| | EGT0001442 | 50 mg | | | | | | | |
| Dose Escalation | EGT0001442 | 5 mg | | | | | | | |
| | EGT0001442 | 10 mg | | | | | | | |
| | EGT0001442 | 20 mg | | | | | | | |
| | EGT0001442 | 50 mg | | | | | | | |

# Listing 16.2.4.3 Prior and Concomitant Medication

| Study<br>Segment | Treatment | Center | Subject<br>Number | ATC Classification<br>WHO Drug Name<br>Medication Name | Start/Stop<br>Date | Ongoing | Drug<br>Strength | Units | Frequency<br>of dose | Route of<br>Administratio | n Indication |
|---|---|---|---|---|---|---|---|---|---|---|---|
| Double-blind | Placebo | 02 | 02141 | ************************************** | ddmmmyyyy,<br>ddmmmyyy | / No | xx | mg | bid | PO | xxxxxxxx |
| Dose Escalation | EGT000144<br>EGT000144<br>EGT000144<br>EGT000144<br>EGT000144<br>EGT000144 | 2 10 mg<br>2 20 mg<br>2 50 mg<br>2 5 mg<br>2 10 mg<br>2 20 mg | 1 | | | | | | | | |

# Listing 16.2.4.4 Inclusion/Exclusion Criteria and Exceptions

| Study | | | Subject | Were all<br>Inclusion/<br>Exclusion | Consent | Washout | Inclusion/Exclusion | | Was a<br>Waiver | Date<br>of Waiver |
|---|---|---|---|---|---|---|---|---|---|---|
| Segment | Treatment | Center | Number | Criteria met? | Date | Type* | Category | No. | Granted? | Granted |
| Double-blind | Placebo | 02 | 02141<br>02142 | Yes<br>No | ddmmmyyyy<br>ddmmmyyyy | | Includion | 2 | Yes | ddmmmyyyy |
| | EGT000144 | 12 5 mg | | | | | | | | |
| | EGT000144 | 12 10 mg | | | | | | | | |
| | EGT000144 | 12 20 mg | | | | | | | | |
| | EGT000144 | 12 50 mg | | | | | | | | |
| Dose Escalation | EGT000144 | 12 5 mg | | | | | | | | |
| | EGT000144 | 12 10 mg | | | | | | | | |
| | EGT000144 | 12 20 mg | | | | | | | | |
| | EGT000144 | 12 50 mg | | | | | | | | |

Note: \*Washout Type: 1 = Diabetic Med Discontinued, 2 = Diabetic Med Naïve

# Listing 16.2.4.5 Urine Drug Screen

| Study<br>Segment | Treatment | Center | Subject<br>Number | Visit<br>Day | Date/Time | Test<br>Name | Test<br>Results |
|---|---|---|---|---|---|---|---|
| Oouble-blind | Placebo | 02 | 02141 | Screening | ddmmmyyyy/hhmm | Amphetamines Barbiturates Cocaine metabolites Opiates Benzodiazepines Cannabinoids Cotinine | Negative |
| | | | | Day 0 | ddmmmyyyy/hhmm | Amphetamines Barbiturates Cocaine metabolites Opiates Benzodiazepines Cannabinoids Cotinine | Negative Negative Negative Negative Negative Negative Negative |
| | EGT000144<br>EGT000144<br>EGT000144<br>EGT000144 | 2 10 mg<br>2 20 mg | | | | | |
| Oose Escalation | EGT000144<br>EGT000144<br>EGT000144 | 2 10 mg<br>2 20 mg | | | | | |

Listing 16.2.5 Study Drug Administration

| Study<br>Segment | Treatment | Center | Subject<br>Number | Dose<br>Day | Did subject fast<br>10 hours<br>Prior to dose? | Dose<br>Date/Time | Dose<br>Status |
|---|---|---|---|---|---|---|---|
| Double-blind | Placebo | 02 | 02141 | 1<br>2<br>3<br>4<br>5<br>6<br>7<br> | Yes<br>Yes<br>Yes | ddmmmyyyy/hhmm | Dosed |
| Dose Escalation | EGT0001442<br>EGT0001442 | 10 mg<br>20 mg<br>50 mg<br>5 mg<br>10 mg<br>20 mg | | | | | |

Listing 16.2.6.1 Fasting Plasma Glucose (mg/dL)

| Study<br>Segment | Treatment | Center | Subject<br>Number | Visit<br>Day | Repeat | Test<br>Date/Time | Observed FPG<br>Results<br>(mg/dL) |
|---|---|---|---|---|---|---|---|
| Double-blind | Placebo | 02 | 02141 | Screening | | ddmmmyyyy/hh:mm | xxxx.x |
| | | | | Day -2 | | ddmmmyyyy/hh:mm | XXXX.X |
| | | | | Day 1 | | ddmmmyyyy/hh:mm | XXXX.X |
| | | | | Day 2 | | ddmmmyyyy/hh:mm | XXXX.X |
| | | | | Day 8 | | ddmmmyyyy/hh:mm | XXXX.X |
| | | | | Day 15 | | ddmmmyyyy/hh:mm | XXXX.X |
| | | | | Day 22 | | ddmmmyyyy/hh:mm | XXXX.X |
| | | | | Day 29 | | ddmmmyyyy/hh:mm | XXXX.X |
| | | | | Day 35 | | ddmmmyyyy/hh:mm | XXXX.X |
| | | | | Day 43 | | ddmmmyyyy/hh:mm | XXXX.X |
| | • • • | | | | | | |
| | EGT0001442 5 mg<br>EGT0001442 10 mg<br>EGT0001442 20 mg<br>EGT0001442 50 mg | | | | | | |
| Dose Escalation | EGT0001442 5 mg | 01 ( | 003 | Screening | | ddmmmyyyy/hh:mm | xxxx.x |
| | 3 | | | Day 0 | | ddmmmyyyy/hh:mm | xxxx.x |
| | | | | Day 1 | | ddmmmyyyy/hh:mm | XXXX.X |
| | | | | Day 2 | | ddmmmyyyy/hh:mm | XXXX.X |
| | | | | Day 3 | | ddmmmyyyy/hh:mm | XXXX.X |
| | | | | Day 8 | | ddmmmyyyy/hh:mm | XXXX.X |
| | | | | Day 15 | | ddmmmyyyy/hh:mm | xxxx.x |
| | | | | Day 22 | | ddmmmyyyy/hh:mm | XXXX.X |
| | | | | Day 29 | | ddmmmyyyy/hh:mm | XXXX.X |
| | | | | Day 43 | | ddmmmyyyy/hh:mm | XXXX.X |
| | EGT0001442 10 mg<br>EGT0001442 20 mg<br>EGT0001442 50 mg | | | | | | |

Listing 16.2.6.2 Weight

| Study<br>Segment | Treatment | Center | Subject<br>Number | Visit<br>Day | Visit<br>Date | Weight<br>(kg) |
|---|---|---|---|---|---|---|
| Double-blind | Placebo | 02 | 02141 | Screening | ddmmmyyyy | XX.X |
| | | | | Day -2 | ddmmmyyyy | xx.x |
| | | | | Day 1 | ddmmmyyyy | XX.X |
| | | | | Day 8 | ddmmmyyyy | XX.X |
| | | | | Day 15 | ddmmmyyyy | xx.x |
| | | | | Day 22 | ddmmmyyyy | XX.X |
| | | | | Day 29 | ddmmmyyyy | xx.x |
| | | | | Day 35 | ddmmmyyyy | xx.x |
| | | | | Day 43 | ddmmmyyyy | xx.x |
| | EGT0001442 10 mg<br>EGT0001442 20 mg<br>EGT0001442 50 mg | | | | | |
| Dose Escalation | EGT0001442 5 mg | 01 | 003 | Screening | ddmmmyyyy | XX.X |
| | - | | | Day 0 | ddmmmyyyy | xx.x |
| | | | | Day 1 | ddmmmyyyy | xx.x |
| | | | | Day 3 | ddmmmyyyy | xx.x |
| | | | | Day 15 | ddmmmyyyy | XX.X |
| | | | | Day 22 | ddmmmyyyy | XX.X |
| | | | | Day 29 | ddmmmyyyy | XX.X |
| | | | | Day 43 | ddmmmyyyy | XX.X |
| | EGT0001442 10 mg<br>EGT0001442 20 mg<br>EGT0001442 50 mg | | | | | |

Dose Escalation EGT0001442 5 mg

# Listing 16.2.6.3 Glycated Hemoglobin A1 (HbA1c) (%)

| Study<br>Segment | Treatment | Center | Subject<br>Number | Visit<br>Day | Repeat | Test<br>Date/Time | Observed HbA1c<br>Results<br>(%) |
|---|---|---|---|---|---|---|---|
| Double-blind | Placebo | 02 | 02141 | Screening<br>Day 1<br>Day 29 | | ddmmmyyyy/hh:mm<br>ddmmmyyyy/hh:mm<br>ddmmmyyyy/hh:mm | xx.x<br>xx.x<br>xx.x |
| | EGT0001442 5 mg EGT0001442 10 mg EGT0001442 20 mg EGT0001442 50 mg | | | | | | |

(Source: path\program name Date/time of run: ddmmmyyyy:hh:mm)

EGT0001442 10 mg EGT0001442 20 mg EGT0001442 50 mg

# Listing 16.2.6.4 24 h UGE (g/day)

| Study<br>Segment | Treatment | Center | Subject<br>Number | Visit<br>Day | Repeat | Test<br>Date/Time | Observed UGE<br>Results<br>(g/day) |
|---|---|---|---|---|---|---|---|
| Double-blind | Placebo | 02 | 02141 | Screening<br>Day 1<br>Day 29 | | ddmmmyyyy/hh:mm<br>ddmmmyyyy/hh:mm<br>ddmmmyyyy/hh:mm | xxxx.x<br>xxxx.x<br>xxxx.x |
| | EGT0001442 5 mg | | | | | | |
| | EGT0001442 10 mg<br>EGT0001442 20 mg<br>EGT0001442 50 mg | | | | | | |
| Dose Escalation | EGT0001442 5 mg<br>EGT0001442 10 mg<br>EGT0001442 20 mg<br>EGT0001442 50 mg | | | | | | |

# Listing 16.2.6.5 Blood (PK) Sample Collection (Dose Escalation Segment)

| Treatment | Center | Subject<br>Number | Sample<br>Number | Study<br>Hour | Scheduled<br>Date | Scheduled<br>Time | Actual<br>Time | Reason for<br>Deviation |
|---|---|---|---|---|---|---|---|---|
| EGT0001442 5 mg | 01 | 003 | 1 | PRE-DOSE | 10Dec2009 | | 0619 | |
| , | | | 2 | 0.5 H | 10Dec2009 | | 0830 | |
| | | | 3 | 1 H | 10Dec2009 | | hhmm | |
| | | | 4 | 2 H | 10Dec2009 | | hhmm | |
| | | | 5 | 3 H | 10Dec2009 | | hhmm | |
| | | | 6 | 4 H | 10Dec2009 | | hhmm | |
| | | | 7 | 6 H | 10Dec2009 | | hhmm | |
| | | | 8 | 8 H | 10Dec2009 | | hhmm | |
| | | | 9 | 10 H | 10Dec2009 | | hhmm | |
| | | | 10 | 12 H | 10Dec2009 | | hhmm | |
| | | | 11 | 24 H | 10Dec2009 | | hhmm | |
| | | | 12 | 48 H | 10Dec2009 | | hhmm | |

EGT0001442 10 mg

EGT0001442 20 mg

EGT0001442 50 mg

Note: Scheduled time is only entered if differ from actual time.

Listing 16.2.6.6 Post Prandial Blood Glucose (mg/dL) (Dose Escalation Segment)

| | | | | | | | Observed | Change fro | |
|---|---|---|---|---|---|---|---|---|---|
| Treatment | Center | Subject<br>Number | | Time<br>Point | Date/Time | Test<br>Name | Results (mg/dL) | Post-meal (mg/dL) | AUC (mg.h/dL) |
| GT0001442 5 mg | 01 | 003 | Day 0 | Prior to Breakfast | 09Dec2009/0845 | BLOOD GLUCOSE | 220 | | |
| | | | | 2 Hours Post Breakfast | 09Dec2009/1107 | BLOOD GLUCOSE | 291 | 71 | |
| | | | | Prior to Lunch | 09Dec2009/1255 | BLOOD GLUCOSE | 176 | | |
| | | | | 2 Hours Post Lunch | 09Dec2009/1517 | BLOOD GLUCOSE | 243 | 67 | |
| | | | | Prior to Dinner | 09Dec2009/1755 | BLOOD GLUCOSE | 184 | | |
| | | | | 2 Hours Post Dinner | 09Dec2009/2018 | BLOOD GLUCOSE | 241 | 57 | |
| | | | | 10:00 PM | 09Dec2009/2245 | BLOOD GLUCOSE | 220 | | xxxx.x |
| | | | Day 2 | Prior to Breakfast | 11Dec2009/0845 | BLOOD GLUCOSE | 220 | | |
| | | | | 2 Hours Post Breakfast | 11Dec2009/1107 | BLOOD GLUCOSE | 272 | 52 | |
| | | | | Prior to Lunch | 11Dec2009/1255 | BLOOD GLUCOSE | 176 | | |
| | | | | 2 Hours Post Lunch | 11Dec2009/1517 | BLOOD GLUCOSE | 243 | 67 | |
| | | | | Prior to Dinner | 11Dec2009/1755 | BLOOD GLUCOSE | 184 | | |
| | | | | 2 Hours Post Dinner | 11Dec2009/2018 | BLOOD GLUCOSE | 243 | 59 | |
| | | | | 10:00 PM | 11Dec2009/2245 | BLOOD GLUCOSE | 220 | | XXXX.X |

. . .

EGT0001442 10 mg

EGT0001442 20 mg

EGT0001442 50 mg

## Listing 16.2.7.1 Treatment Emergent Adverse Events

| | | System Organ Class | | | | | | | Relationship | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Study<br>Segment | Treatment | Contor | Subject | | Preferred Term Verbatim Term | | solution<br>Time | | Severity# | to<br>Study Drug¹ | Action<br>Taken² | Outcome |
| | | Center | Nullber | NO. | verbatim ieim | | | serious:~ | severity# | Study Drug- | | |
| Double-blind | Placebo | 02 | 02141 | 1 | ************************************** | ddmmmyyyy<br>ddmmmyyyy | | 0 | 1 | 2 | 0 | 1 |
| | | | • • • | | | | | | | | | |
| | | 1442 5 | _ | | | | | | | | | |
| | | 1442 10 | _ | | | | | | | | | |
| | | 1442 20 | _ | | | | | | | | | |
| | EGTOOO | 1442 50 | ) mg | | | | | | | | | |
| Dose Escalatio | n EGT000 | 1442 5 | mg | | | | | | | | | |
| | EGT000 | 1442 10 | ) mg | | | | | | | | | |
| | EGT000 | 1442 20 | ) mg | | | | | | | | | |
| | EGT000 | 1442 50 | ) ma | | | | | | | | | |

Note: \* Serious?: 1 = Yes, 2 = No

Sorting by: Study segment, Treatment, Center, Subject, Start Date, Start Time, End Date, End Time

<sup>#</sup> Severity: 1 = Mild, 2 = Moderate, 3 = Severe.

<sup>1</sup> Relationship to study drug: 1 = Yes, 2 = No

<sup>&</sup>lt;sup>2</sup> Action taken: 1 = None, 2 = Medication Administered, 3 = Non-Drug Therapy, 4 = Hospitalization, 5 = Discontinuation From Study, 6 = Other.

<sup>&</sup>lt;sup>3</sup> Outcome: 1= Resolved, 2 = Continuing with Treatment, 4 = Continuing without Treatment, 10 = Death.

# Similar Listings:

Listing 16.2.7.2 Drug-related Treatment Emergent Adverse Events

Listing 16.2.7.3 Serious Treatment Emergent Adverse Events

Listing 16.2.7.4 Treatment Emergent Adverse Events Leading to Study Discontinuation

Listing 16.2.7.5 Cardiovascular Treatment Emergent Adverse Events

### Listing 16.2.7.6 Pre-treatment Adverse Events

| Study<br>Segment | Center | Subject<br>Number | AE<br>No. | System Organ Class<br>Preferred Term<br>Verbatim Term | Onset/Resolution<br>Date Time | Serious?* | Severity# | Relationship<br>to<br>Study Drug <sup>1</sup> | Action<br>Taken <sup>2</sup> | Outcome <sup>3</sup> |
|---|---|---|---|---|---|---|---|---|---|---|
| Double-blind | 02 | 02141 | 1 | ************************************** | ddmmmyyyy hh:mm/<br>ddmmmyyyy hh:mm | | 1 | 2 | 0 | 1 |

. . .

Dose Escalation

#### Note:

- \* Serious?: 1 = Yes, 2 = No
- # Severity: 1 = Mild, 2 = Moderate, 3 = Severe.
- 1 Relationship to study drug: 1 = Yes, 2 = No
- <sup>2</sup> Action taken: 1 = None, 2 = Medication Administered, 3 = Non-Drug Therapy, 4 = Hospitalization, 5 = Discontinuation From Study, 6 = Other.
- <sup>3</sup> Outcome: 1= Resolved, 2 = Continuing with Treatment, 4 = Continuing without Treatment, 10 = Death.

Sorting by: Study segment, Washout type, Center, Subject, Start Date, Start Time, End Date, End Time

#### Listing 16.2.7.7 Adverse Events during Washout Period

| | | | | | System Organ Class | | | | | Relationship | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Study<br>Segment | Washou | | Subject<br>Number | AE<br>No. | Preferred Term Verbatim Term | Onset/Res | solution<br>Time | Serious?* | Severitv# | to<br>Study Drug¹ | Action<br>Taken² | Outcome <sup>3</sup> |
| | | Center | | NO. | verbacim leim | | | Jerrous: | | | | |
| Double-blind | 1 | 02 | 02141 | 1 | xxxxxxxxxxxxx<br>xxxxxxxxxxx<br>xxxxxxxxxx | ddmmmyyyy<br>ddmmmyyyy | | 0 | 1 | 2 | 0 | 1 |

Dose Escalation

Note: + Washout type: 1= Diabetic Med Discontinued, 2= Diabetic Med Naive

- \* Serious?: 1 = Yes, 2 = No
- # Severity: 1 = Mild, 2 = Moderate, 3 = Severe.
- <sup>1</sup> Relationship to study drug: 1 = Yes, 2 = No
- <sup>2</sup> Action taken: 1 = None, 2 = Medication Administered, 3 = Non-Drug Therapy, 4 = Hospitalization, 5 = Discontinuation From Study, 6 = Other.
- <sup>3</sup> Outcome: 1= Resolved, 2 = Continuing with Treatment, 4 = Continuing without Treatment, 10 = Death.

Sorting by: Study segment, Washout type, Center, Subject, Start Date, Start Time, End Date, End Time

# Listing 16.2.8.1 Clinical Laboratory Test Results in Biochemistry

| | | | | | | Lab | | | S: | I Uni | t | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Study | | | Subjec | t Age/ | Visit | | | Lab | Test | | Normal | | |
| - | Treatment | Center | _ | _ | Day Repeat | Date | Time | | Results | Unit | | Flag * | Comments |
| Double-blind | Placebo | 02 | 02141 | 36/M | Screening | ddmmmyyy | y hh:mm | Albumin<br>Calcium<br>Creatini | | XX<br>XX<br>XX | xx-xx<br>xx-xx | L(NCS) | xxxxxxxx |
| Dose Escalation | EGT0001442 5 mg EGT0001442 10 r EGT0001442 20 r EGT0001442 50 r EGT0001442 5 mg EGT0001442 10 r EGT0001442 20 r | mg<br>mg | | | | | | | | | | | |

Note: \* Flag: L = Low, H = High, NCS = Not clinical significance, CS = Clinical significance

Table will continue for other biochemistry lab tests.

# Similar listings:

Listing 16.2.8.2 Clinical Laboratory Test Results in Hematology

Listing 16.2.8.3 Clinical Laboratory Test Results in Urinalysis

Listing 16.2.8.4 Vital Signs

| Study<br>Segment | Treatment | Center | Subject<br>Number | Visit<br>Day | Seated for 5 minutes? | Heart<br>Rate<br>(BPM) | Systolic<br>BP<br>(mmHg) | Diastolic<br>BP<br>(mmHg) | Respiratory<br>Rate<br>(breaths/min) | Temperature |
|---|---|---|---|---|---|---|---|---|---|---|
| Double-blind | Placebo | 02 | 02141 | Screening | Yes | xxx | xxx | xxx | XX.X | xx.x |
| | | | | Day -2 | Yes | XXX | XXX | XXX | XX.X | XX.X |
| | | | | Day 1/Pre-dose | Yes | XXX | XXX | XXX | XX.X | XX.X |
| | | | | Day 2/Pre-dose | Yes | XXX | XXX | XXX | XX.X | XX.X |
| | | | | Day 8 | Yes | XXX | XXX | XXX | XX.X | XX.X |
| | | | | Day 15 | Yes | XXX | XXX | XXX | XX.X | XX.X |
| | | | | Day 22 | Yes | XXX | XXX | XXX | XX.X | XX.X |
| | | | | Day 29 | Yes | XXX | XXX | XXX | XX.X | XX.X |
| | | | | Day 35 | Yes | XXX | XXX | XXX | XX.X | XX.X |
| | | | | Day 43 | Yes | XXX | xxx | xxx | xx.x | xx.x |
| | EGT0001442 10<br>EGT0001442 20<br>EGT0001442 50 | mg | | | | | | | | |
| Dose Escalation | EGT0001442 5 | mg 01 | 003 | Screening | Yes | xxx | XXX | XXX | XX.X | XX.X |
| | | | | Day 0 | Yes | XXX | XXX | XXX | XX.X | XX.X |
| | | | | Day 1/Pre-dose | Yes | XXX | XXX | XXX | XX.X | XX.X |
| | | | | Day 1/1 hr | Yes | XXX | XXX | XXX | XX.X | XX.X |
| | | | | Day 1/2 hr | Yes | XXX | XXX | XXX | XX.X | XX.X |
| | | | | Day 1/4 hr | Yes | XXX | XXX | XXX | XX.X | XX.X |
| | | | | Day 1/8 hr | Yes | XXX | XXX | XXX | XX.X | XX.X |
| | | | | Day 2/Pre-dose | Yes | XXX | XXX | XXX | XX.X | XX.X |
| | | | | Day 3/Pre-dose | Yes | XXX | XXX | XXX | XX.X | XX.X |
| | | | | Day 8 | Yes | XXX | XXX | XXX | XX.X | XX.X |
| | | | | Day 15 | Yes | XXX | XXX | XXX | XX.X | XX.X |
| | | | | Day 22 | Yes | XXX | XXX | XXX | XX.X | XX.X |
| | | | | Day 29 | Yes | XXX | XXX | XXX | XX.X | XX.X |
| | | | | Day 43 | Yes | XXX | xxx | XXX | XX.X | xx.x |
| | EGT0001442 10<br>EGT0001442 20<br>EGT0001442 50 | mg | | | | | | | | |

# Listing 16.2.8.5 12-Lead ECG

| Study<br>Segment | Treatment | Center | Subject<br>Number | | Ventri<br>cular<br>Rate<br>(BPM) | PR | QRS<br>Interval<br>(ms) | QT<br>Interval<br>(ms) | QTc<br>Interval<br>(ms) | ECG<br>Findings<br>(NCS/CS) | | t ECG<br>s Description |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Double-blind | Placebo | 02 | 02141 | Screening Day -2 Day 1/Pre-dose Day 2/Pre-dose Day 29 | xxx<br>xxx<br>xxx<br>xxx | XXX<br>XXX<br>XXX | XXX<br>XXX<br>XXX | XXX<br>XXX<br>XXX | XXX<br>XXX<br>XXX | Normal<br>Abnormal (NCS)<br>Normal<br>Normal | ) NR | xxxxxx |
| | EGT0001442 5 n<br>EGT0001442 10<br>EGT0001442 20<br>EGT0001442 50 | mg<br>mg | | | | | | | | | | |
| Dose Escalation | EGT0001442 5 n | mg 01 | 003 | Screening Day 0 Day 1/Pre-dose Day 1/ 2 hr Day 2/Pre-dose Day 29 | xxx<br>xxx<br>xxx<br>xxx<br>xxx | XXX<br>XXX<br>XXX<br>XXX | XXX<br>XXX<br>XXX<br>XXX | XXX<br>XXX<br>XXX<br>XXX | xxx<br>xxx<br>xxx | Normal<br>Normal<br>Normal<br>Normal<br>Normal | | |
| | EGT0001442 10<br>EGT0001442 20<br>EGT0001442 50 | mg | | | | | | | | | | |

Note:

CS = Clinically Significant
NCS = Not Clinically Significant

# Listing 16.2.8.6 Self Monitored Blood Glucose (SMBG)

| Study<br>Segment | Treatment Ce | enter | Subject<br>Number | Visit<br>Day | Date | Time | Results<br>(mg/dL) |
|---|---|---|---|---|---|---|---|
| Double-blind | Placebo 02 | ) | 02141 | DAY-14 | ddmmmyyyy | HHMM | xxx |
| | | | | DAY-13 | ddmmmyyyy | HHMM | XXX |
| | | | | DAY-12 | ddmmmyyyy | HHMM | XXX |
| | | | | DAY-11 | ddmmmyyyy | HHMM | xxx |
| | | | | DAY-10 | ddmmmyyyy | HHMM | xxx |
| | | | | DAY-9 | ddmmmyyyy | HHMM | xxx |
| | | | | DAY-8 | ddmmmyyyy | HHMM | xxx |
| | | | | DAY-7 | ddmmmyyyy | HHMM | xxx |
| | | | | DAY-6 | ddmmmyyyy | HHMM | xxx |
| | | | | DAY-5 | ddmmmyyyy | HHMM | xxx |
| | | | | DAY-4 | ddmmmyyyy | HHMM | XXX |
| | | | | DAY-3 | ddmmmyyyy | HHMM | xxx |
| | | | | DAY-2 | ddmmmyyyy | HHMM | XXX |
| | | | | DAY-1 | ddmmmyyyy | HHMM | XXX |
| | | | | DAY 0 | ddmmmyyyy | HHMM | XXX |
| | | | | DAY 1 | ddmmmyyyy | HHMM | XXX |
| | | | | DAY 2 | ddmmmyyyy | UNK | XXX |
| | | | | DAY 3 | ddmmmyyyy | UNK | XXX |
| | | | | Day 43 | ddmmmyyyy | HHMM | XXX |
| | EGT0001442 5 | | | | | | |
| | EGT0001442 10<br>EGT0001442 20 | _ | | | | | |
| | EGT0001442 20 | _ | | | | | |
| Dose Escalation | EGT0001442 5 | | | | | | |
| | EGT0001442 10 | ) mg | | | | | |
| | EGT0001442 20 | ) mg | | | | | |
| | EGT0001442 50 | ) ma | | | | | |

Note: SMBG are measured daily after washout starts till the last termination visit.

Note: table will continue for other Days.

### Listing 16.2.8.7 Physical Examination

| Study<br>Segment | Treatment | Center | Subject<br>Number | Visit<br>Day | Change<br>from<br>Previous | Body<br>System | Examination<br>Finding |
|---|---|---|---|---|---|---|---|
| Double-blind | Placebo | 02 | 02141 | Screening | | Skin Head Eyes Ears Nose Throat Neck Thyroid Lungs Heart Abdomen Lymph Nodes Extremities | Sunburn left hand (peeling skin) Normal |
| | | | | Day -2 | Yes | Skin | Normal |
| | EGT0001442 | 5 ma | | | | | |
| | EGT0001442<br>EGT0001442<br>EGT0001442 | 10 mg<br>20 mg | | | | | |
| Dose Escalation | EGT0001442<br>EGT0001442<br>EGT0001442<br>EGT0001442 | 10 mg<br>20 mg | | | | | |

Note: table will continue for Days 1,8,15,22,29,35 and 43 for double-blind segment. table will continue for screening, Days 0,1,3,8,15,22,29 and 43 for dose escalation segment.

# **Figures**

Figure 14.2.1 Fasting Plasma Glucose (mean± SE) - Double-blind Segment



Figure 14.2.2 Fasting Plasma Glucose in Change from Baseline (mean± SE) - Double-blind Segment



Note: Baseline is defined as the mean of FPG values on day -2 and day 1.

Similar Figures:

Figure 14.2.3 Body Weight (mean± SE) - Double-blind Segment

Figure 14.2.4 Body Weight in Change from Baseline (mean± SE) - Double-blind Segment

Figure 14.2.5 HbA1c (mean± SE) - Double-blind Segment



Figure 14.2.6 24h UGE (mean± SE) - Double-blind Segment



Figure 14.2.7 Mean Plasma Concentration for EGT0001442 (ng/mL) - Dose Escalation Segment



Similar Figures:

Figure 14.2.8 Individual Plasma Concentration for EGT0001442 (ng/mL) - Dose Escalation Segment